#### **CONFIDENTIAL**

#### The GlaxoSmithKline group of companies

208832

: Worldwide Development

Division

Information Type : Reporting and Analysis Plan (RAP)

Title : A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics and Tolerability of Cabotegravir and Rilpivirine Long-Acting Injections Following Intramuscular Administration in the Vastus Lateralis Muscle of Healthy Adult Participants

Compound Number : GSK1265744

Effective Date : 07-MAY-2021

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 208832
- This RAP is intended to describe the safety, pharmacokinetics, and tolerability analyses required for the study
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## The GlaxoSmithKline group of companies

## **RAP Author(s):**

| Author | Date |
|------------------------------------------------------|-------------|
| Lead | |
| PPD | 07 MAN 2021 |
| Statistician (HIV, GSK Clinical Statistics) | 07-MAY-2021 |
| <b>Co-Authors</b> | |
| PPD | 07-MAY-2021 |
| Principal Programmer (HIV, GSK Clinical Programming) | |

## **RAP Team Review Confirmations:** (Method: E-mail)

| Reviewer | Date |
|----------------------------------------------------------|-------------|
| PPD | 07-MAY-2021 |
| Clinical Development Manager (R&D GCSD, GSK) | |
| PPD | 06-MAY-2021 |
| Principal Clinical Data Manager (GCDO, GSK Clinical Data | |
| Management) | |
| PPD | 06-MAY-2021 |
| Manager, Clinical Pharmacology (GSK CPMS) | |
| PPD | 06-MAY-2021 |
| PPD , Research & Development (ViiV | |
| Healthcare) | |

# Clinical Statistics & Clinical Programming Line Approvals: (Method: Pharma TMF eSignature)

| Approver | Date |
|------------------------------------------------------|-------------|
| PPD | 05-MAY-2021 |
| Statistics Leader (HIV, GSK Clinical Statistics) | |
| PPD | 07-MAY-2021 |
| Programming Director (HIV, GSK Clinical Programming) | |

Copyright 2021 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| 1. | REPORTING & ANALYSIS PLAN SYNOPSIS | 5 |
| | 1.1. Revision Chronology | 5 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 6 |
| | 2.1. Changes to the Protocol Defined Statistical Analysis Plan | 6 |
| | 2.2. Study Objective(s) and Endpoint(s) | |
| | 2.3. Study Design | 8 |
| | 2.4. Statistical Hypotheses | |
| | 2.4.1. Hypotheses | |
| 3. | PLANNED ANALYSES | 9 |
| ٠. | 3.1. Interim Analyses | |
| | 3.2. Final Analyses | |
| 4. | ANALYSIS POPULATIONS | 10 |
| 4. | 4.1. Protocol Deviations | |
| | 4.1. Protocol Deviations | 11 |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONVENTIONS | |
| | 5.1. Treatment and Other Sub-Group Descriptions for Data Displays | |
| | 5.2. Baseline Definitions | 13 |
| | 5.3. Other Considerations for Data Analyses and Data Handling | |
| | Conventions | |
| | 5.3.1. Other Considerations | 13 |
| 6. | STUDY POPULATION | 15 |
| | 6.1. Subject Disposition | 15 |
| | 6.2. Demographic and Baseline Characteristics | 15 |
| | 6.3. Medical History and Concomitant Medications | |
| 7. | SAFETY ANALYSES | 15 |
| ٠. | 7.1. Extent of Exposure and Treatment Compliance | |
| | 7.2. Adverse Events | |
| | 7.3. Injection Site Reaction Adverse Events | |
| | 7.4. Adverse Events of Special Interest (AESIs) | 17 |
| | 7.5. Pregnancies (as applicable) | |
| | 7.6. Clinical Laboratory Evaluations | |
| | 7.7. Other Safety Analyses | |
| 0 | DUADAM COMMETIC ANALYCES | 40 |
| 8. | PHARMACOKINETIC ANALYSES | |
| | 8.1. Drug Concentration Measures | |
| | 8.2. Deriving and Summarizing Pharmacokinetic Parameters | |
| | 8.3. Statistical Analyses | |
| | 8.4. Strategy for Intercurrent Events – Covid-19 Complications | 20 |
| 9. | HEALTH OUTCOMES ANALYSES | 21 |
| | 9.1. CCI | |
| | 9.2. | 21 |

## CONFIDENTIAL

| 10. | REFE | RENCES. | | 22 |
|---|---|---|---|---|
| 11 | ΔPPFI | NDICIES | | 23 |
| | 11.1. | | x 1: Schedule of Activities | |
| | 11.1. | | Screening and Oral Lead-in Phase | |
| | | | CAB LA + RPV LA Injection Phase and Follow- up | |
| | 11.2. | 11.1.Z. | x 2: Assessment Windows | 20<br>27 |
| | 11.2. | | Definitions of Assessment Windows | |
| | 11 2 | | | 21 |
| | 11.3. | Appendix | x 3: Study Phases and Treatment Emergent Adverse | 20 |
| | | 11.3.1. | Study Phases | |
| | 44.4 | 11.3.2. | | 30 |
| | 11.4. | | x 4: Data Display Standards and Handling Conventions | 31 |
| | | 11.4.1. | Reporting Process | |
| | | 11.4.2. | Reporting Standards | |
| | | 11.4.3. | Reporting Standards for Pharmacokinetic Data | 32 |
| | | 11.4.4. | Reporting Standards for Liver Safety Data | 32 |
| | | | 11.4.4.1. Liver Stopping/Monitoring Criteria | |
| | | | 11.4.4.2. Hepatobiliary Abnormality Criteria | 33 |
| | 11.5. | | x 5: Derived and Transformed Data | |
| | | 11.5.1. | General | |
| | | 11.5.2. | Study Population | |
| | | 11.5.3. | Safety | |
| | | 11.5.4. | Pharmacokinetic | 37 |
| | | 11.5.5. | Health Outcomes | 37 |
| | 11.6. | Appendix | x 6: Reporting Standards for Missing Data | 39 |
| | | | Premature Withdrawals | |
| | | 11.6.2. | Handling of Missing Data | 39 |
| | | | 11.6.2.1. Handling of Missing and Partial Dates | |
| | 11.7. | Appendix | x 7: Values of Potential Clinical Importance | 41 |
| | | 11.7.1. | Laboratory Values | |
| | | 11.7.2. | • | |
| | 11.8. | | x 8: Abbreviations & Trademarks | |
| | | | Abbreviations | |
| | | | Trademarks | |
| | 11.9. | | x 9: List of Data Displays | |
| | 11.0. | 11.9.1. | Data Display Numbering | |
| | | 11.9.2. | Deliverables | |
| | | 11.9.3. | Study Population Tables | |
| | | 11.9.4. | Safety Tables | |
| | | 11.9.5. | Safety Figures | |
| | | 11.9.6. | Pharmacokinetic Tables | |
| | | 11.9.0. | Pharmacokinetic Figures | |
| | | - | 9 | |
| | | 11.9.8. | Health Outcomes Tables | |
| | | 11.9.9. | ICH Listings | |
| | | | Non-ICH Listings | |
| | 44.40 | | Mock Displays | |
| | 11.10. | • • | x 10: AESI Identification | |
| | | | Hepatotoxicity | |
| | | | Seizures | |
| | | 11.10.3. | Torsade de pointes/QT prolongation | 75 |
| | | 11.10.4. | COVID-19 Adverse Events | 76 |

## 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Pharmacology Study Report for Protocol 208832. |
| Protocol | This RAP is based on the original protocol (Dated 02-MAR-2020) of study GSK1265744/208832 (GSK Document No.: 2018N357118_00) and its protocol amendment 1 (Dated 13-AUG-2020; GSK Document No.: 2018N357118_01) |
| Primary<br>Objective | To describe the PK profiles of CAB and RPV following a single intramuscular injection each of CAB LA + RPV LA administered to the lateral thigh muscle in adult healthy participants |
| Primary<br>Endpoint | <ul> <li>Maximum observed concentration (C<sub>max</sub>) and time of maximum observed concentration (t<sub>max</sub>) in plasma</li> <li>Area under the concentration – time curve from time zero to last quantifiable time point (AUC<sub>0-t</sub>) through the follow-up phase</li> <li>Area under the concentration – time curve from time zero to infinity (AUC<sub>0-∞</sub>)</li> <li>Apparent terminal phase half-life (t½) and absorption rate constant (K<sub>A</sub>LA)</li> </ul> |
| Study<br>Design | This is a Phase 1, open label study conducted in healthy participants to assess the PK of CAB and RPV in plasma following a single 600 mg (1 x 3 mL) and a 900 mg (1 x 3 mL) injection each, respectively, administered IM to separate <i>vastus lateralis</i> muscles on each leg. The study will consist of a 30-day screening phase, a 28-day oral lead-in (OLI) phase at a CAB dose of 30 mg and RPV dose of 25 mg once a day with a meal, followed by a 10-14 day washout phase. Single doses of CAB and RPV will then be injected, administered IM: 600 mg (1 x 3 mL) CAB on left and a 900 mg (1 x 3 mL) RPV injection on right <i>vastus lateralis</i> muscles. Sparse PK sampling for up to 29 days in OLI and serial PK sampling for up to 4 weeks after the injection, per SoA. Participants will return for safety assessments and additional PK sampling at Week 8, 12, 24, 36, and 52 post last injection during the follow-up phase. |
| Planned<br>Analyses | All the derived PK parameters will be listed and summarized by treatment and study phase. For each of these PK parameters the following descriptive summary statistics will be calculated: n, arithmetic mean with associated 95% CI, standard deviation, median, minimum, and maximum. The mean & geometric mean with associated 95% CIs, standard deviations, and geometric coefficient of variation (CV <sub>b</sub> (%)) will be calculated for all parameters except t <sub>tmax</sub> . |
| Analysis Populations | Enrolled Population, Safety Population, Pharmacokinetic Concentration Population and Pharmacokinetic Parameter Population |
| Hypothesis | No formal hypothesis will be tested in this study |
| Primary<br>Analyses | Primary endpoints include CAB and RPV PK parameters $C_{max}$ , $AUC_{0-t}$ , $AUC_{0-\infty}$ , $t_{1/2}$ , and $K_ALA$ as calculated from injection phase concentration-time data. Descriptive statistics and graphics will be created to describe the primary PK endpoints of interest. |

## 1.1. Revision Chronology

| Revision Chronology: | | |
|----------------------|-------------|---------------------|
| ID: 35421_2099331 | 31-AUG-2020 | Critical Components |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

Cabotegravir (CAB) is an integrase inhibitor being developed in combination with rilpivirine (RPV, TMC278), a non-nucleoside reverse transcriptase inhibitor, for the treatment of HIV. CAB is currently in Phase 3 development as monotherapy for the prevention of sexually-acquired HIV-1 infection. CAB and RPV are separately formulated as oral tablets for once daily administration and as long-acting (LA) aqueous suspensions for parenteral administration monthly or every 2-months. RPV 25mg oral tablets is approved as EDURANT in multiple countries, including the USA, Europe and Canada, for use in antiretroviral (ARV) treatment-naïve patients.

A two-drug long-acting, monthly antiretroviral regimen of CAB + RPV has demonstrated good efficacy, tolerability, and long-term safety in HIV-infected adults following oral and monthly and every 2-month IM dosing in the gluteus muscle for durations exceeding 3 years in Phase 2 and Phase 3 studies [LATTE; LATTE-2; ATLAS, 2019; FLAIR, 2019, ATLAS-2M]. Review and approval of the CAB + RPV regimen for treatment of HIV infection is ongoing.

Separate early Phase 1 studies of CAB LA and RPV LA evaluated PK and tolerability of single and repeat-dose injections in other anatomic locations including abdomen (subcutaneous) and IM administration in the ventrogluteal muscle (CAB), gluteus maximus muscle (RPV), and deltoid muscle (RPV) in healthy volunteers [HIV Therapy 2013; International AIDS Society 2013; RPV LA NATAP report]. Gluteal injections of CAB LA + RPV LA were progressed in late-stage studies given better participant tolerability to injections at this injection site with the anticipated injection dosing volume required to achieve desired exposures.

There remains considerable interest in exploring alternative injection sites either as an alternative rotational (e.g. gluteal injection fatigue) or chronic injection site (e.g. gluteal implants contraindicating injection or young pediatric populations without sufficient gluteal mass for injection). The *vastus lateralis* muscle in the thigh has been used as an injection location for other drugs (e.g. epinephrine, etc.) and is a common injection site in young children (e.g. vaccines). Moreover, self- or partner-injection of CAB LA + RPV LA in the thigh muscle may be explored in future studies pending favorable pharmacokinetics, safety, and tolerability of CAB LA + RPV LA thigh injections.

The objective of this study is to evaluate the pharmacokinetics, tolerability, and safety of CAB LA + RPV LA administered concomitantly as two separate IM injections in the *vastus lateralis* muscle of adult healthy participants. Data from this study will be used to inform the feasibility of administering CAB LA + RPV LA in the *vastus lateralis* muscle in HIV-infected children <12 years of age and adult populations.

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

In consideration of the recent, global Covid-19 pandemic, and in accordance with recent GSK clinical guidance, sensitivity analyses summarizing disposition and select safety results will be displayed alongside primary results. This stands as an addition to the originally planned statistical analysis specified in the protocol dated 02-MAR-2020 and

protocol amendment 1 dated 13-AUG-2020. A second addition will be the calculation of PK parameters in the OLI phase alongside the PK parameters of the Injection phase as noted in the primary objective. Thirdly, the protocol calls for the short version questionnaire to be implemented while this RAP plans for the full version, administered separately for each thigh, in order to collect clinically meaningful information on the future use of thigh injections in the pediatric population. Finally, listings are specified to be inclusive of all screened subjects.

Changes from the originally planned statistical analysis specified in the protocol and its amendment 1 are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | Rationale |
|---|---|---|
| Study objectives and endpoints<br>listed without consideration of the<br>Covid-19 pandemic | Disposition and select safety<br>results will be repeated with<br>consideration to subjects'<br>relation to Covid-19. | The Covid-19 pandemic<br>has spurred the need to<br>assess whether the<br>impact creates substantial<br>impact on study results. |
| PK parameters only calculated for Injection phase | Applicable PK parameters will<br>also be calculated in the OLI<br>phase as data permits | OLI PK parameters are of<br>interest in addition to<br>Injection parameters |
| Short version of column questionnaire recorded | Full version of the column questionnaire recorded separately for each injection | Information found in the full version is considered clinically meaningful to plan for further thigh injections in children. |
| PK Listings are subset by population relevant to the data | All listing data will be shown<br>for all screened subjects | To more feasibly serve as<br>a reference for subjects<br>not meeting population<br>requirements |

## 2.2. Study Objective(s) and Endpoint(s)

Table 2 Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To describe the PK profiles of CAB and RPV following a single intramuscular injection each of CAB LA + RPV LA administered to the lateral thigh muscle in adult healthy participants. | <ul> <li>Maximum observed concentration (C<sub>max</sub>) and time of maximum observed concentration (t<sub>max</sub>) in plasma</li> <li>Area under the concentration – time curve from time zero to last quantifiable time point (AUC<sub>0-t</sub>) through the follow-up phase</li> <li>Area under the concentration – time curve from time zero to infinity (AUC<sub>0-∞</sub>)</li> <li>Apparent terminal phase half-life (t½) and absorption rate constant (K<sub>A</sub>LA)</li> </ul> |

| Safety Objectives | Safety Endpoints |
|---|---|
| To assess safety and tolerability of<br>CAB and RPV following repeated oral<br>dose and single intramuscular injection<br>in the lateral thigh of healthy<br>participants | Safety and tolerability parameters including<br>adverse events (AEs), clinical laboratory tests,<br>electrocardiogram (ECG), and vital sign<br>assessments |
| Secondary Objectives | Secondary Endpoints |
| To assess liver safety and tolerability<br>of CAB and RPV following repeated<br>oral dose and single intramuscular<br>injection in the lateral thigh of adult<br>healthy participants | Tolerability parameters (liver related adverse events) and liver chemistry abnormalities |
| <b>Exploratory Objectives</b> | Exploratory Endpoints |

# CCI Exploratory Enapoints

## 2.3. Study Design

This is a phase 1, open label study in healthy participants to assess the PK of CAB and RPV in plasma following a single 600 mg (1 x 3 mL) and a 900 mg (1 x 3 mL) injection each; respectively, administered IM to separate *vastus lateralis* muscles on each leg.

The study will consist of

- 30-day screening period
- 28-day oral lead-in (OLI) phase at a CAB dose of 30 mg and RPV dose of 25 mg once a day with a meal
- 10 14 days washout period
- CAB and RPV injection, administered IM: 600 mg (1 x 3 mL) CAB on left and a 900 mg (1 x 3 mL) RPV injection on right *vastus lateralis* muscle
- Sparse PK sampling for up to 29 days in OLI and serial PK sampling for up to 4 weeks after the injection, per SoA. Participants will return for safety assessments and additional PK sampling at Week 8, 12, 24, 36, and 52 post last injection during the follow-up phase.

Approximately 15 adult healthy participants will be dosed with injectable study interventions. If participants prematurely discontinue the study, for any other reason,

other than an AE, additional replacement participants may be enrolled at the discretion of the Sponsor in consultation with the investigator. The study design is defined in Table 3.

Table 3 Study Design

| Screening | Oral<br>Lead-in | Washout | CAB Injection and Compartmental PK Sampling | Safety/<br>Blood Plasma Sampling |
|---|---|---|---|---|
| Within 30 days<br>of Oral Lead-in | | No drug<br>administered 10 -<br>14 days | Single 600 mg CAB LA IM dose into lateral thigh + single 900 mg RPV LA IM dose into opposite lateral thigh | |
| | x 28 days | | Serial blood plasma sampling up to 4 weeks post-injection | 52 Weeks post-dose |

Figure 1 Study Schematic



Injection Day 1: CAB LA 600mg IM (3mL) + RPV LA 900mg IM (3mL) Lateral thigh

## 2.4. Statistical Hypotheses

## 2.4.1. Hypotheses

The primary objective of this study is to describe the PK profiles of CAB and RPV following a single intramuscular injection each of CAB LA + RPV LA administered to the lateral thigh muscle. No formal statistical hypotheses are to be tested. Where appropriate, an estimation approach will be taken, and point estimates and confidence intervals will be constructed. There will be no formal comparison.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

There will be no formal interim analysis. All preliminary safety, tolerability and available pharmacokinetic data may be reviewed internally at any time point. Depending on feasibility, evaluation of PK data may be performed at time points such as Week 4 and Week 12 post injection for preliminary PK analysis.

## 3.2. Final Analyses

Final analysis will be performed after all subjects have completed the study and final database freeze (DBF) has been declared by Data Management. Data will be listed and summarized according to GSK reporting standards, where applicable.

Statistical data analyses will be performed by, or under the direct auspices of, Clinical Statistics and Programming, GlaxoSmithKline utilizing SAS version 9.4 or higher. PK analysis of the plasma CAB and RPV concentration-time data will be conducted using non-compartmental methods with WinNonlin (Version 6.3 or higher).

All the derived PK parameters will be listed and summarized by treatment and study phase. For each of these PK parameters the following descriptive summary statistics will be calculated: n, arithmetic mean with associated 95% CI, standard deviation, median, minimum, and maximum. The mean & geometric mean with associated 95% CIs, standard deviations, and geometric coefficient of variation ( $CV_b(\%)$ ) will also be calculated for all parameters except  $t_{max}$ .

Safety and health outcome data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards.

#### 4. ANALYSIS POPULATIONS

As a convention, listing data will be displayed for all screened subjects.

Table 4 Study Populations

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Enrolled | <ul> <li>All participants who sign the ICF.</li> <li>Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Study Population |
| Safety | All participants who take at least 1 dose of study drug. | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic<br>Concentration<br>(PC) | All participants who undergo plasma PK sampling and<br>have evaluable PK assay results from either oral or<br>injection dosing | <ul> <li>Concentration<br/>summaries</li> <li>Individual plotting<br/>of concentration-<br/>time data</li> </ul> |
| Pharmacokinetic Parameter (PP) | <ul> <li>All participants who undergo plasma PK sampling and have evaluable PK parameters estimated.</li> <li>Note: PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded.</li> </ul> | <ul> <li>PK parameter<br/>summaries</li> <li>Mean/median plots<br/>and summary<br/>tables</li> </ul> |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, excluded medications, conduct of the trial, participant management, or participant assessment) will be summarized with frequencies and proportions by study phase and overall.

Protocol deviations will be tracked by the study team throughout the conduct of the study.

- Data will be reviewed prior to freezing the database to ensure all significant deviations and deviations which may lead to exclusion from the analysis populations are captured and categorized on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

All protocol deviations will be listed. A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Treatment and Other Sub-Group Descriptions for Data Displays

Data display treatment descriptors with actual treatment dose will be defined as displayed in Table 5. Safety events in the washout phase will be counted with events in the Oral lead-in phase. Safety events in the Follow-up phase will be counted separately from the Injection phase.

Table 5Study Treatment

| | | Treatment Group Descriptions | | | |
|---|---|---|---|---|---|
| Phase | Analysis | Data Set | | Final Data Display (i.e. HARP / other) | |
| | | Code | Treatment<br>Description | Treatment Description- Footnote | Column Header |
| Oral Lead-in | PK | A | Oral CAB 30mg<br>tablet once daily x<br>4 weeks lead-in | Oral CAB<br>30mg=Cabotegravi<br>r 30mg PO 4<br>weeks lead-in | Oral CAB 30mg |
| | | В | Oral RPV 25mg<br>tablet once daily x<br>4 weeks lead-in | Oral RPV 25mg=<br>Rilpivirine 25mg<br>PO 4 weeks lead-<br>in. | Oral RPV 25mg |
| | Safety | AB | Oral CAB 30mg +<br>RPV 25mg tablets<br>once daily x 4<br>weeks lead-in | Oral CAB 30mg + Oral RPV 25mg =Cabotegravir 30mg + Rilpivirine 25mg PO 4 weeks lead-in | Oral CAB 30mg +<br>Oral RPV 25mg |
| Injection, PK, Safety (ISRs), HO | | С | Single 600mg CAB<br>LA IM dose | IM CAB<br>600mg=Cabotegra<br>vir IM 600mg<br>single dose. | IM CAB 600mg –<br>Injection Phase;<br>IM CAB 600mg –<br>Follow-up Phase |
| | | D | Single 900mg RPV<br>LA IM dose | IM RPV<br>900mg=Rilpivirine<br>IM 900mg single<br>dose. | IM RPV 900mg –<br>Injection Phase;<br>IM RPV 900mg –<br>Follow-up Phase |
| | Safety | CD | Single 600mg CAB<br>+ single 900mg<br>RPV LA IM dose | IM CAB 600mg + IM RPV 900mg = Cabotegravir IM 600mg + Rilpivirine IM 900mg single dose. | IM CAB 600mg + IM RPV 900mg - Injection Phase; IM CAB 600mg + IM RPV 900mg - Follow-up Phase |

#### 5.2. Baseline Definitions

For safety parameters the baseline or pre-dose value will be the latest assessment prior to the time of study drug administration in each phase with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and considered for use as baseline. If there are multiple assessments collected on the same scheduled time, the average of these assessments will be used. Table 6 indicates the baseline day to be used in the analysis.

Table 6 Baseline Parameter Specifications

| Phase | Parameter | Study Assessments Considered as<br>Baseline | Baseline Used in Data<br>Display |
|---|---|---|---|
| Oral Lead-in Phase | Laboratory results,<br>Vital Sign results,<br>ECG results <sup>1</sup> | OLI Baseline = last non-missing pre-dose<br>assessment collected <= Date of first OLI<br>dose | OLI Day 1 |
| Injection Phase | Laboratory results, Vital Sign results (pre-dose), ECG results¹ (pre-dose), scores | Injection Phase Baseline = assessment collected on the date of CAB + RPV injection | Injection Day 1 |
| Follow-up Phase | Laboratory results,<br>Vital Sign results<br>(pre-dose), ECG<br>results¹ (pre-dose) | Follow-up Phase Baseline = assessment collected on the date of CAB + RPV injection | Injection Day 1 |

<sup>1.</sup> Average of the triplicate assessments for quantitative assessments will be used as the baseline.

If time is not collected, Day 1 assessments are assumed to be taken prior to first dose of the respective phase. Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

#### 5.3.1. Other Considerations

Other considerations for data analyses, including information regarding premature withdrawal, unscheduled assessments, derived and transformed data, and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.1 | Appendix 1: Schedule of Activities |
| 11.2 | Appendix 2: Assessment Windows |
| 11.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 11.4 | Appendix 4: Data Display Standards and Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Reporting Standards for Missing Data |

## CONFIDENTIAL

## 

| Section | Component |
|---------|-----------------------------------------------------|
| 11.7 | Appendix 7: Values of Potential Clinical Importance |
| 11.8 | Appendix 8: Abbreviations & Trademarks |
| 11.9 | Appendix 9: List of Data Displays |
| 11.10 | Appendix 10: AESI Identification |

## 6. STUDY POPULATION

The study population analyses will be based on both the Enrolled and Safety populations, unless otherwise specified.

Study population analyses include analyses of study populations, subjects' disposition, important protocol deviations, demographic and baseline characteristics, and prior and concomitant medications. Outputs will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

## 6.1. Subject Disposition

A summary table will be generated to provide the count of subjects included in each analysis population for the study (see Section 4 for definition of analysis populations).

The End of Study Record will be summarized by study phase and overall. Counts for the all discontinuation categories will be repeated considering subjects who discontinued to a Covid-19 related incident.

A disposition listing will include whether subjects prematurely withdrew from the study, the reason for premature discontinuation along with the start and end date of investigational product (IP) dosing and the date of completion or premature discontinuation from the study. An additional listing showing subjects who discontinued to Covid-19 considerations will be included.

## 6.2. Demographic and Baseline Characteristics

Demographic data include date of birth, sex, race, and ethnicity. Demographic data and baseline characteristics (i.e. height, weight, and BMI) will be summarized for the Safety Population. Race will be further summarized separately from the other demographic characteristics. All demographic data will be listed by subject.

## 6.3. Medical History and Concomitant Medications

Medical history events will be summarized and listed. Concurrent medication verbatim text will be coded and classified by the Anatomical Therapeutic Chemical Classification level 1 (ATC Level 1) code and the preferred term using the GSK coding system, GSK DRUG. Concomitant medications will then be summarized by ATC classification, study phase, and overall. Coding of concurrent medications will be the responsibility of the GSK coding group.

## 7. SAFETY ANALYSES

Safety data will be summarised and listed by, or under the direct auspices of, Clinical Statistics, GlaxoSmithKline. The safety summaries will be based on the Safety population, unless otherwise specified and shown for the Oral Lead-in, Injection, and Follow-up phases where applicable.

Safety endpoints include:

- Safety and tolerability parameters including adverse events, clinical laboratory tests, ECG, and vital sign assessments
- Tolerability parameters (liver related adverse events) and liver chemistry abnormalities

For continuous safety parameters, the Injection phase Baseline will also serve as Follow-up phase Baseline. No formal statistical analysis of the safety data will be conducted. The precise format and content of Safety tables and listings are shown in Appendix 9 of the RAP.

## 7.1. Extent of Exposure and Treatment Compliance

Overall CAB & RPV exposure will be presented with descriptive statistics (i.e. n, mean, SD, median, minimum, and maximum) by study phase and treatment. Treatment will be determined by the laterality of the injection. CAB will be administered on a subject's *left* thigh while RPV will be administered on a subject's *right* thigh. Parameters displayed will include number of days of oral exposure, oral compliance percentage, and injection status. Details on oral compliance percentage calculation are included in Appendix 5.

A by-subject listing of data on subject exposure will be generated including dose date and time, unit, formulation, route, frequency and location.

#### 7.2. Adverse Events

Adverse event verbatim text will be coded and classified by system organ class (body system) and preferred term using a standardized GSK coding system: Medical Dictionary for Regulatory Activities (MedDRA, v23.0 or higher). AE data will be summarized with frequencies and percent by study phase and overall. The relationship of AE system organ class, preferred term, and verbatim text will be listed. Treatment emergent AEs, drugrelated AEs, serious adverse events (SAEs) including fatal AEs, and AEs leading to drug withdrawal or study discontinuation will be summarized by study phase and overall. AEs and drug-related AEs will also be summarized by maximum toxicity grade (based on Division of AIDS (DAIDS) categories). All AEs will be listed by subject and AE start date.

Adverse events related to Covid-19 will also be summarized by SOC, PT, and maximum toxicity. Subjects with Covid-19 tests performed as well as Covid-19 diagnoses will also be summarized. Summaries of serious Covid-19 AEs and Covid-19 AEs leading to study discontinuation or drug withdrawal will also be presented in accordance with Covid-19 safety assessment guidance. Covid-19 AEs will also be presented by sex and pandemic course (during and post-) if applicable.

## 7.3. Injection Site Reaction Adverse Events

Injection site reaction adverse event data will also be summarized by treatment and overall. Tables will include subject and event-level summaries. ISR treatment will be determined by the laterality of the assessment (left vs. right). All ISR AEs will be shown in a separate listing from overall adverse events.

## 7.4. Adverse Events of Special Interest (AESIs)

AESIs will be summarized for Hepatotoxicity and Seizures. QT Prolongation events will be listed. A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event for Adverse Events of Special Interest (AESI). [Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting.] The details of the current planned grouping, including Standardized MedDRA Query (SMQ) values (as applicable), and planned displays are provided in Appendix 10: AESI Identification and Appendix 9: List of Data Displays.

## 7.5. Pregnancies (as applicable)

If any female subjects become pregnant during the study, a listing of such subjects will be provided.

## 7.6. Clinical Laboratory Evaluations

Worst grade post-baseline for hematology, clinical chemistry, and urinalysis data will be summarized by study phase. Summaries of change from baseline in hematology and clinical chemistry by study phase and visit will be created. If any laboratory test results are outside of the reference range, they will be flagged with high/low and/or toxicity grade in the listing. Standardized units will be used for clinical laboratory summary tables and listings.

Hematology, clinical chemistry, drug, infectious disease, coagulation and urinalysis data will be listed by subject, study phase, visit, and collection date.

## 7.7. Other Safety Analyses

Vital sign data (temperature, systolic and diastolic blood pressure, and pulse rate) will be summarized by study phase, visit, and planned time. Absolute values and change from baseline values will be shown. Injection phase Baseline will also serve as Follow-up phase Baseline. Vitals signs will be listed by subject, study phase, visit, planned time, and actual date and time.

Electrocardiogram (ECG) data including values and findings will be summarized by study phase, visit, and timepoint. Absolute values and change from baseline will be shown for PR, QRS, QT, QTcB, and QTcF results. Baseline will be calculated as the mean of triplicate readings recorded prior to first dose in each study phase.

All ECG data including clinical interpretation will be listed by subject, study phase, visit and record date. Clinically significant ECG abnormalities will be flagged and listed separately, and corresponding values will be provided.

Liver related adverse events and chemistry abnormalities will be summarized separately by study phase. See Appendix 10 for a list of Hepatotoxicity AEs and Appendix 7 for Chemistry values of Potential Clinical Importance.

## 8. PHARMACOKINETIC ANALYSES

The reconciliation of the PK Case Report Form (CRF) and SMS2000 data will be performed by, or under the direct auspices of, Clinical Pharmacology Sciences and Study Operations (CPSSO), GlaxoSmithKline.

The merge of PK concentration data and CRF data will be performed by, or under the direct auspices of, Clinical Statistics (Programmer), GlaxoSmithKline.

Derivation of pharmacokinetic parameters will be performed by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline.

Statistical analysis of pharmacokinetic parameters will be performed by, or under the direct auspices of, Clinical Statistics (Statistician), GlaxoSmithKline.

Concentration and PK parameter data will be reported for specified Pharmacokinetic populations in the OLI and Injection phases.

## 8.1. Drug Concentration Measures

Plasma CAB and RPV concentration values will be summarized with descriptive statistics by study phase, treatment, visit, and planned timepoint for the PK Concentration Population (PC). These concentration values will be determined directly from concentration-time data from each analyte. Descriptive statistics including the n, mean with associated 95% CI, standard deviation, median, minimum, maximum, geometric mean with associated 95% CI, standard deviation of logarithmically transformed data,  $5^{th}/95^{th}$  percentiles and the geometric coefficient of variation ( $CV_b(\%)$ )).

Individual concentration-time profiles and median/mean profiles from each analyte in each study phase will be plotted for the PK Concentration (PC) Population. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. semi-log plot). Actual assessment times will be used in the individual concentration-time plots. Nominal times will be used for the purposes of summarization and in mean and median plots. See Appendix 4: Data Display Standards & Handling Conventions. for details on pharmacokinetic figure and table displays.

## 8.2. Deriving and Summarizing Pharmacokinetic Parameters

Pharmacokinetic parameters will be derived by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 6.3 or higher (Pharsight, Inc., Cary, NC). All calculations of non-compartmental PK parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits. The following PK parameters will be derived and displayed for the PP Population as data permits:

Table 7 Derived PK Parameters

| Parameter | Parameter Description | OLI Phase | Injection Phase |
|---|---|---|---|
| C <sub>max</sub> | Maximum observed concentration | Day 1 | Overall |
| t <sub>max</sub> | Time of occurrence of C <sub>max</sub> | Day 1 | Overall |
| AUC <sub>0</sub> -∞ | Area under the concentration time curve from time zero to infinity | Day 1-2 | Overall |
| AUC <sub>0-t</sub> | Area under the concentration time curve from time zero to last quantifiable time point | Day 1-2 | Overall |
| t <sub>1/2</sub> | Terminal phase half-life | Day 1-2 | Overall |
| K <sub>A</sub> LA | Absorption rate constant, Long-acting | NA | Overall |
| λz | Terminal phase rate constant | Day 1-2 | NA |
| C24 | Concentration at OLI Phase 24-hour timepoint | Day 2 | NA |
| Сτ | Trough concentrations (Cτ) at OLI Phase Day 29 | Day 29 | NA |

NOTES: NA: Not Applicable

Primary Pharmacokinetic endpoints include the following PK parameters from Injection Phase:

- Maximum observed concentration (Cmax) and time of maximum observed concentration (t<sub>max</sub>) in plasma
- Area under the concentration time curve from time zero to last quantifiable time point (AUC<sub>0-t</sub>) through the follow-up phase
- Area under the concentration time curve from time zero to infinity (AUC<sub>0- $\infty$ </sub>)
- Apparent terminal phase half-life ( $t\frac{1}{2}$ ) and absorption rate constant ( $K_ALA$ ))

PK parameters such as  $C_{max}$  and AUC should be reported in  $\mu g/mL$  and  $\mu g^*h/mL$  for CAB and in ng/mL and  $ng^*h/mL$  for RPV. Other PK parameters such as  $t_{max}$  and  $t_{1/2}$  should be reported in hours and  $K_ALA$  and  $\lambda z$  parameters in /h for both CAB and RPV.

Additional parameters may be included as required.

## 8.3. Statistical Analyses

All the derived pharmacokinetic parameters will be summarized and listed for the PP population by study phase and treatment. For each of these PK parameters, with the exception of  $t_{max}$ , the following descriptive summary statistics will be calculated for each treatment: n, arithmetic mean with associated 95% CI, standard deviation, median, minimum, maximum, geometric mean with associated 95% CI, standard deviation of logarithmically transformed data, and the geometric coefficient of variation (CV<sub>b</sub>(%)). For  $t_{max}$ , the n, median, minimum, and maximum summary statistics will be provided.

Data display specifications for derived PK parameter summaries and listings are given in Appendix 9 of this RAP

PK samples collected outside the protocol defined time-windows and/or other protocol deviations will be reviewed by the study team to determine whether the sample will be excluded from PK analyses. PK reporting will also consider planned Quality Tolerance Limit (QTL) outcomes affecting study data quality. Details are found in the QTL Report.

## 8.4. Strategy for Intercurrent Events – Covid-19 Complications

While incidents of Covid-19 could be expected to affect subject safety, its effect on CAB + RPV PK concentrations is unknown. Given the small study sample size implying less likelihood that a subject acquires Covid-19 through the course of the study, the benefit of a sensitivity analysis for subjects that acquire Covid-19 during the course of their PK sampling appears minimal. Should more information become available and/or the clinical need arise, this RAP may be amended to include Covid-19 PK sensitivity analyses in order to further understand any potential interacting effects.

## 9. HEALTH OUTCOMES ANALYSES

Health outcomes questionnaire data will be summarised and listed by, or under the direct auspices of, Clinical Statistics, GlaxoSmithKline. The health outcomes analyses will be based on the Safety population, unless otherwise specified. All questionnaire data will be listed by subject, item, treatment, and timepoint as applicable.

No formal statistical analysis of the health outcomes data will be conducted. The precise format and content of health outcomes tables and listings are shown in Appendix 5 of the RAP.



## 10. REFERENCES

GlaxoSmithKline Document Number 2018N357118\_00: A Phase 1, Multicompartment Pharmacokinetic Study of Cabotegravir Long-acting in Healthy Adult Volunteers. Effective Date: 02-MAR-2020

GlaxoSmithKline Document Number 2018N357118\_01: A Phase 1, Multicompartment Pharmacokinetic Study of Cabotegravir Long-acting in Healthy Adult Volunteers. Effective Date: 13-AUG-2020

GlaxoSmithKline Document: Covid-19 Guidance for Estimands and Estimation.

GlaxoSmithKline Document: Impact of Covid-19 on Assessment of Safety in Clinical Trials.

## 11. APPENDICIES

## 11.1. Appendix 1: Schedule of Activities

## 11.1.1. Screening and Oral Lead-in Phase

| Study Period | Screening <sup>1</sup> | | | Oral Lead-ii | 1 <sup>9</sup> | Day 29 | Early<br>Withdrawal <sup>9</sup> | Washout Period |
|---|---|---|---|---|---|---|---|---|
| | 3 | | Do | sing Days ' | 1-28 | ] | | |
| Visit Window | Within<br>30 days<br>of oral lead-in | Day -1 | Day 1 | Day 2 | Day 14 | Within 24 hours<br>of the Day 28 last<br>dose | EW | 10 – 14 days |
| Informed Consent | Χ | | | | | | | |
| Demographics | Х | | | | | | | |
| Medical / Medication / Drug /<br>Alcohol History | Х | | | | | | | |
| Inclusion/Exclusion Criteria <sup>2</sup> | Х | | Х | | | | | |
| Height, Weight, BMI | Х | | | | | | | |
| Physical Exam | Х | | Х | | | | | |
| Vital Signs <sup>3</sup> | Х | | Х | Х | Х | Х | Х | |
| 12-Lead ECG | Х | | Х | | | X | | |
| Drug / Alcohol Screen <sup>3</sup> | Х | | Х | | | | | |
| Pregnancy Test <sup>3</sup> | Х | | Х | | Χ | Х | | |
| Testing for SARS-CoV-24 | Х | Χ | | | | | | |
| Hepatitis B, Hepatitis C Screening | Х | | | | | | | |
| HIV Test | Х | | | | | | | |
| Urine Dipstick | Х | | | | | | | |
| Hematology with differential;<br>Clinical Chemistry Tests <sup>3</sup> | Х | | Х | Х | Х | Х | X | |
| Coagulation Tests | Х | | | | | | | |
| Admit to clinic | | Х | | | | | | |
| Dispense Oral lead-in IP | | | Х | | | | | |

| Study Period | Screening <sup>1</sup> | | | Oral Lead-ii | n <sup>9</sup> | Day 29 | Early<br>Withdrawal <sup>9</sup> | Washout Period |
|---|---|---|---|---|---|---|---|---|
| | | | Do | sing Days | 1-28 | 1 -1.7 -1 | | |
| Visit Window | Within<br>30 days<br>of oral lead-in | Day -1 | Day 1 | Day 2 | Day 14 | Within 24 hours<br>of the Day 28 last<br>dose | EW | 10 – 14 days |
| Administer oral CAB + RPV <sup>5</sup> | | | X | Х | Х | | | |
| Dispense Medication Dosing Diary | | | | Х | | | | |
| Drug accountability/ pill count/review drug diary | | | | Х | Х | Х | | |
| Blood plasma PK sampling <sup>6</sup> | | | Х | Х | Х | Х | Х | |
| AE Assessment <sup>7</sup> | | | Х | Х | Х | X | Χ | |
| Concomitant Medication Review | | | Х | Х | Х | X | Х | |
| Genetic sample <sup>8</sup> | | | Х | | | | | |
| Discharge from the clinic | | _ | | Х | | | | |

- 1. Screening may occur over more than one visit but within 30 days of the first dose of oral CAB and RPV in the oral lead in phase.
- 2. Eligibility criteria must be carefully assessed at the Screening visit and confirmed at the Day 1 Oral lead-in phase visit and re-confirmed prior to injection.
- 3. Prior to administering the first oral dose of CAB and RPV, study personnel must verify the following pre-dose assessments to be within normal limits prior to administration: vital signs, pregnancy test (negative; Females of Reproductive Potential (FRP) only. The results of the Drug/Alcohol screen, hematology with differential, and clinical chemistry tests on Day 1 are not required prior to administering the first oral doses of CAB and RPV but should be drawn prior to CAB and RPV administration.
- 4. Following the second test for SARS-CoV-2, participants will be advised to self-quarantine until entrance to the unit while awaiting final testing clearance.
- 5. Oral CAB and RPV dosing Days 1 to 28. Day 1, Day 2, and Day 14 doses should be administered in the clinic.
- 6. PK sampling On Day 1 1h, 2h, 3h, 4h, 6h, 8h, and 12h, and Day 2 PK between 22-26 h from first oral dose. On Day 14 pre-dose samples. Day 29 assessments should occur between 22-26 hours from the last dose on Day 28. Total of 20 PK samples (10 for CAB, 10 for RPV assay) will be collected during oral lead-in phase. Please refer to Protocol Section 8.4 for permitted PK window for OLI phase.
- 7. AE assessment will include a brief, symptom-directed physical exam as needed.
- 8. Genetic sample collect the sample at the earliest convenient time after the first dose in the oral lead in phase on Day 1.
- 9. If a participant is withdrawn prior to receiving the CAB LA and/or RPV LA injection, a follow-up/withdrawal visit should be scheduled 10-14 days after the last oral dose of CAB and RPV.

## 11.1.2. CAB LA + RPV LA Injection Phase and Follow- up

| | | Injection Phase | | | | | | | Follow-up | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | lı | njectio<br>Day 1 | n | Day 2 | Day 4 | Day 5 | Day 7/8 | Day 10 | Day 15 | Day 17 | Day 22 | Day 28<br>(Week 4) | Week 8 | Week 12 | Week 24 | Week 36 | Week 52 | Withdrawal <sup>1</sup> |
| | Pre-<br>dose <sup>2</sup> | 1h | 2h | 24h | 72h | 96h | 168h | | | | | | | | | | | |
| Permitted window for PK collection | Within 1 h prior to dosing | ± 15 min | ± 30 min | ±2h | ±2h | ±2h | ±2h | ±2h | ±2h | ±2h | ± 2 h | ±2h | ± 3 days | ± 3 days | ± 3 days | ± 3 days | ±3 days | |
| Interim Medical/Medication/<br>Drug / Alcohol History <sup>2</sup> | Х | | | | | | | | | | | | | | | | | |
| Pregnancy Test | Х | | | | | | | | | | | Χ | Х | Χ | Χ | Χ | Χ | Х |
| 12-Lead ECG <sup>2</sup> | Х | | Χ | | | Χ | | | | | | | | | | | Χ | Х |
| HIV Test | Х | | | | | | | | | | | | | | Х | | Χ | Х |
| Testing for SARS-CoV-2 | | | | | | | | | | | | | | | | | | |
| Hematology; Clinical Chemistry | Χ | | | | | | Χ | | | Χ | | Х | Χ | Χ | Χ | Χ | Χ | Χ |
| Vital Signs <sup>2</sup> | Χ | | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ |
| Administer CAB LA + RPV LA <sup>2</sup> | Χ | | | | | | | | | | | | | | | | | |
| CCI | | X3 | | X3 | X3 | X3 | X <sup>3</sup> | | | | | | | | | | | |
| Injection site reaction assessment | | Х | Х | X | Х | Х | X | Х | X | X | Х | X | Х | Х | X | X | Х | Х |
| AE Assessment <sup>4</sup> | | Х | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ |
| Concomitant Medication Review | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | Х |
| Blood plasma PK Sampling <sup>5</sup> | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Х | Χ |

#### **CONFIDENTIAL**

208832

- 1. Participants who terminate before week 52 will be asked to return to the site for a withdrawal visit.
- 2. On Day 1, study personnel must verify the following pre-dose assessments to be within normal limits prior to injection: ECG, vital signs, pregnancy test (negative; FRP only), review AE assessment, and concomitant medications. If a clinical abnormality, clinically significant AE, or prohibited medication that precludes injection is observed/recorded, the medical monitor must be contacted for further instruction.
- 3. Participants will be asked to describe the comfort level with the injections received.
- 4. AE assessment will include a brief, symptom-directed physical exam as needed.
- 5. Total of 34 PK samples (17 each for CAB and RPV) will be collected through CAB LA + RPV LA Injection Phase and Follow-up.

## 11.2. Appendix 2: Assessment Windows

All assessments/events (including those from planned, unscheduled and withdrawal visits) will be assigned to assessment windows/analysis visits according to actual dates of collection rather than the nominal visit labels recorded on the eCRF or in the laboratory database. All assessment data, including unscheduled data will be presented in listings.

For parameters which are not scheduled to be assessed at a particular visit, the all-inclusive assessment windows will still be used; however, data displays summarizing measurements by visit will only report visits in which the parameter is a planned collection according to Appendix 1: Schedule of Activities

Note: Prior to visit slotting, assessments are first assigned to a study phase according to Table 3.

#### 11.2.1. Definitions of Assessment Windows

Table 8 Assessment Windows for Screening and OLI Phase Data

| Parameter | Analysis Window | Target<br>Period Day | Analysis<br>Timepoint |
|---|---|---|---|
| Assess | sments assigned to Phase=Screening or OLI (p | per <u>Table 3</u> ) | |
| All | OLI Phase Day <1 | The day of earliest record | Screening |
| PK, Vital Signs, Labs, ECG | OLI Phase Day = 1 | 1 | Day 1 |
| PK, Vital Signs, Labs | OLI Period Day = 2 | 2 | Day 2 |
| PK | 13 ≤ OLI Phase Day ≤ 15 | 14 | Day 14 |
| Vital Signs, Labs | 3 ≤ OLI Phase Day ≤ 21 | 14 | Day 14 |
| PK | 28 ≤ OLI Phase Day ≤ 30 | 29 | Day 29 |
| Vital Signs, Labs, ECG | 22 ≤ OLI Phase Day | 29 | Day 29 |
| | If none of the above | | |

Table 9 Assessment Windows for Injection & Follow-up Phase Data

| Parameter <sup>a</sup> | Analysis Window | Target<br>Period | Analysis<br>Timepoint |
|---|---|---|---|
| | | Day | ' |
| Assessm | ents assigned to Phase=Injection (per | Table 3) | |
| PK, Vital Signs, Labs, ECG, | Injection Phase Day = 1 | 1 | Day 1 |
| PK, Vital Signs, | Injection Phase Day = 2 | 2 | Day 2 |
| PK | Injection Phase Day = 4 | 4 | Day 4 |
| CCI | 3 ≤ Injection Phase Day ≤ 4 | 4 | Day 4 |
| PK | Injection Phase Day = 5 | 5 | Day 5 |
| Vital Signs | 3 ≤ Injection Phase Day ≤ 6 | 5 | Day 5 |
| CCI | 5 ≤ Injection Phase Day ≤ 6 | 5 | Day 5 |
| ECG | 2 ≤ Injection Phase Day | 5 | Day 5 |

| Parameter <sup>a</sup> | Analysis Window | Target<br>Period<br>Day | Analysis<br>Timepoint |
|---|---|---|---|
| PK | Injection Phase Day = 7 | 7 | Day 7 |
| PK | Injection Phase Day = 8 | 8 | Day 8 |
| CCI | 7 ≤ Injection Phase Day | 8 | Day 8 |
| Vital Signs | 7 ≤ Injection Phase Day ≤ 9 | 8 | Day 8 |
| Labs | 2 ≤ Injection Phase Day ≤ 10 | 8 | Day 8 |
| PK | Injection Phase Day = 10 | 10 | Day 10 |
| Vitals | 10 ≤ Injection Phase Day ≤ 12 | 10 | Day 10 |
| PK | Injection Phase Day = 15 | 14 | Day 15 |
| Vital Signs | 12 ≤ Injection Phase Day ≤ 16 | 14 | Day 15 |
| PK | Injection Phase Day = 17 | 17 | Day 17 |
| Vital Signs | 17 ≤ Injection Phase Day ≤ 19 | 17 | Day 17 |
| Labs | 11 ≤ Injection Phase Day ≤ 23 | 17 | Day 17 |
| PK | Injection Phase Day = 22 | 22 | Day 22 |
| Vital Signs | 20 ≤ Injection Phase Day ≤ 25 | 22 | Day 22 |
| PK | Injection Phase Day = 28 | 28 | Week 4 |
| Vital Signs | 26 ≤ Injection Phase Day | 28 | Week 4 |
| Labs | 24 ≤ Injection Phase Day | 28 | Week 4 |
| | If none of the above | | Day X, where<br>X=Injection Phase<br>Day |
| Ass | sessments assigned to Phase=Follow-up (per | Table 3) | |
| Vital Signs, Labs | (Date of Nominal Follow-up Week 4<br>Visit – CAB + RPV Injection Date) +2<br>≤ Injection Phase Day ≤ 70 | 56 | Week 8 |
| PK | 53 ≤ Follow-up Period Day ≤ 59 | 56 | Week 8 |
| Vital Signs, Labs | 71 ≤ Follow-up Period Day ≤ 126 | 84 | Week 12 |
| PK | 81 ≤ Follow-up Period Day ≤ 87 | 84 | Week 12 |
| Vital Signs, Labs | 127 ≤ Follow-up Period Day ≤ 210 | 168 | Week 24 |
| PK | 165 ≤ Follow-up Period Day ≤ 171 | 168 | Week 24 |
| Vital Signs, Labs | 211 ≤ Follow-up Period Day ≤ 308 | 252 | Week 36 |
| PK | 249 ≤ Follow-up Period Day ≤ 255 | 252 | Week 36 |
| Vital Signs, Labs, ECG | 309 ≤ Follow-up Period Day | 364 | Week 52 |
| PK | 361 ≤ Follow-up Period Day ≤ 367 | 364 | Week 52 |
| | If none of the above | | Day X, where<br>X=Follow-up<br>Phase Day |
| NOTES: OLI Day, Injection Day, and | d Follow-up Day are defined in Section 11.5.1. | | |

# 11.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

## 11.3.1. Study Phases

All assessments and events (including those collected as planned, early withdrawal and unscheduled visits) will be classified in study phases according to <u>Table 3</u>.

Assessments/events are assigned to study phases sequentially, starting from the top of each table.

 Table 3
 Assignment of Study Phases

| For All Events or | Assessments |
|---|---|
| Study Period | Date range |
| Screen | If actual "Time of Day" for the assessment/event is collected: |
| | Start Date and Time < OLI Treatment Start Date & Time |
| | If actual "Time of Day" for the assessment/event is not collected: |
| | Start Date < OLI Treatment Start Date |
| OLI Phase | If actual "Time of Day" for the assessment/event is collected: |
| | For participants continuing into Injection Phase: OLI Treatment Start Date & Time ≤ Start Date & Time < Date & Time of CAB + RPV Injection |
| | For participants not continuing into Injection Phase: OLI Treatment Start Date & Time |
| | If actual "Time of Day" for the assessment/event is not collected: |
| | For participants continuing into Injection Phase: OLI Treatment Start Date ≤ Start Date < Date of CAB + RPV Injection |
| | For participants not continuing into Injection Phase: OLI Treatment Start Date ≤ Start Date |
| Injection Phase | If actual "Time of Day" for the assessment/event is collected: |
| | Date & Time of CAB + RPV Injection ≤ <b>Start Date &amp; Time</b> and <b>Start Date</b> ≤ Date of Nominal Follow-up Week 4 |
| | If actual "Time of Day" for the assessment/event is not collected: |
| | Date of CAB + RPV Injection ≤ <b>Start Date</b> ≤ Date of Nominal Follow-up Week 4 Visit |
| Follow-up Phase | Date of Nominal Follow-up Week 4 Visit < Start Date |

#### NOTES:

Date = Date of assessment

## **Table 4** Study Phases for Concomitant Medication

| Concomitant during: | |
|---|---|
| Study Period | Date range |
| Prior | Medication Taken < OLI Treatment Start Date & Time |
| OLI Phase | For participants continuing into Injection Phase: OLI Treatment Start Date & Time ≤ Medication Taken < Injection Phase Treatment Start Date & Time |
| | For participants not continuing into Injection Phase: OLI Treatment Start Date & Time ≤ Medication Taken |
| Injection Phase | Injection Phase Treatment Start Date & Time ≤ <b>Medication Taken</b> ≤ Date of Nominal Follow-up Week 4 Visit |
| Follow-Up Phase | Date of Nominal Follow-up Week 4 Visit < Medication Taken |

#### NOTES:

- If concomitant medication time is missing, the medication will be assumed to be taken predose, prior to that day's treatment dosing.
- Please refer to Appendix 6: Reporting Standards for Missing Data. for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 11.3.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | AEs will be considered emergent in the OLI, Injection and Follow-up Phases according to the classification defined in <a href="Table 3">Table 3</a> . AEs that occur in the Follow-up Phase will be considered Treatment Emergent. |

## 11.4. Appendix 4: Data Display Standards and Handling Conventions

## 11.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software version 9.4 will be used. | |
| Reporting Area | |
| HARP Server | us1salx00259 |
| HARP Compound | \ARPROD\GSK1265744\mid213199\internal_01 |
| \ARPROD\GSK1265744\mid213199\internal_02 | |
| | \ARPROD\GSK1265744\mid213199\primary_01 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.1.</li> </ul> | |
| Generation of RTF Files | |
| <ul> <li>RTF files will be generated for all tables in Appendix 9: List of Data Displays.</li> </ul> | |

#### 11.4.2. Reporting Standards

#### General

 The current GSK Statistical Display Standards in the GSK Standards Library (IDSL) will be applied for reporting, unless otherwise stated (Library Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK Statistical Display Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting
  of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the GSK Standard Statistical Display Principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any important deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to GSK Standard Statistical Display Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using assessment windows defined in Section 11.2.1.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Schedule of Activities in Section 11.1).
- Evaluable assessments at unscheduled visits will be used when categorizing values across visits, such as 'maximum grade during the injection phase'.

| Descriptive Summary Statistics |
|---|
| Continuous Data Refer to GSK Standard Statistical Display Principle 6.06.1 |
| Categorical Data N, n, frequency, % |
| Graphical Displays |
| Refer to GSK Standard Statistical Display Principals 7.01 to 7.13. |

#### 11.4.3. **Reporting Standards for Pharmacokinetic Data**

| Pharmacokinetic Concentration Data Descriptive Summary Statistics, Graphical Displays and Listings Refer to IDSL Statistical Principle 6.06.1. For continuous data: Not quantifiable values (NQs) at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood. For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration); for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present) for summary statistics, these are set to 0 (to avoid skewing of the summary statistics) Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly). If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing). Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only | | |
|---|---|---|
| Refer to IDSL Statistical Principle 6.06.1. For continuous data: Not quantifiable values (NQs) at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood. For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration); for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present) for summary statistics, these are set to 0 (to avoid skewing of the summary statistics) Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly). If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing). Note: Concentration values will be imputed as per GUI_51487 for descriptive summary | Pharmacokinetic Cond | centration Data |
| Statistics/arialysis and sammanized graphical displays smy. | Descriptive Summary<br>Statistics, Graphical | <ul> <li>Refer to IDSL PK Display Standards.</li> <li>Refer to IDSL Statistical Principle 6.06.1.</li> <li>For continuous data: <ul> <li>Not quantifiable values (NQs) at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood.</li> <li>For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration);</li> <li>for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present)</li> <li>for summary statistics, these are set to 0 (to avoid skewing of the summary statistics)</li> </ul> </li> <li>Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly).</li> <li>If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing).</li> </ul> |

**Reporting Standards for Liver Safety Data** 

## 11.4.4.1. **Liver Stopping/Monitoring Criteria**

11.4.4.

| Element | Reporting Detail |
|---|---|
| General | A liver monitoring event occurs when subject meets predefined liver chemistry monitoring criteria that trigger increased monitoring of the subject's liver chemistries, |
| | but no action is taken with study treatment unless liver chemistry stopping criteria are |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>met. A liver stopping event occurs when subject meets predefined liver chemistry stopping criteria, ALT &gt;=3xULN for this study, that trigger discontinuation of study treatment and requirement of additional actions and follow up assessments to be performed. For subjects with more than one liver stopping or liver monitoring event, only data related to the earliest most severe criteria event is included in displays.</li> <li>Resolved is defined as ALT &lt;3xULN for 2 consecutive visits or &lt;3xULN for one visit if subject discontinued and no data available. Post treatment records are included to evaluate resolution of the event.</li> </ul> |

## 11.4.4.2. Hepatobiliary Abnormality Criteria

| Element | Reporting Detail |
|---|---|
| General | To include ALT, ALP, Bilirubin, & INR parameters |
| ALT >=3xULN and BIL >=2xULN | <ul> <li>If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be &gt;=35% when total bilirubin is &gt;=2xULN, in order to satisfy the criteria.</li> <li>Bilirubin value is on or up to 28 days after ALT value.</li> </ul> |
| ALT >=3xULN and INR >1.5 | INR value is on or up to 28 days after ALT value. |
| ALT >=3xULN and BIL >=2xULN and ALP 2 (<1%) <2xULN | <ul> <li>If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be &gt;=35% when total bilirubin is &gt;=2xULN, in order to satisfy the criteria.</li> <li>Bilirubin value is on or up to 28 days after ALT value.</li> <li>The ALP value must occur on or up to 28 days after the ALT value.</li> </ul> |
| Hepatocellular injury | Hepatocellular injury is defined as ((ALT/ALT ULN)/(ALP/ALP ULN)) >=5 and ALT >=3xULN. ALT and ALP values must occur on the same day. |
| Hepatocellular injury and BIL >=2xULN | <ul> <li>Hepatocellular injury is defined as ((ALT/ALT ULN)/(ALP/ALP ULN)) &gt;= 5 and ALT &gt;= 3xULN. ALT and ALP values must occur on the same day.</li> <li>If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be &gt;= 35% when total bilirubin is &gt;= 2xULN, in order to satisfy the criteria.</li> <li>Bilirubin value is on or up to 28 days after ALT value.</li> </ul> |
| BIL >=2xULN | If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be >=35% when total bilirubin is >=2xULN, in order to satisfy the criteria. |
| AST >3xULN and ALP <2xULN and BIL >=2xULN | <ul> <li>ALP and BIL values must occur on or up to 28 days after AST value.</li> <li>If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be &gt;=35% when total bilirubin is &gt;=2xULN, in order to satisfy the criteria.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| ALT>=X ULN and AST>=X ULN | <ul> <li>AST and ALT values must occur on the same day</li> </ul> |

## 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- If there are multiple measurements within a time window (per Section 11.2.1), the value closest to the
  target day for that window will be used. If values are the same distance from the target, then the mean of
  the measurements (for quantitative parameters including ECG values) or the worst-case of the
  measurements (for qualitative parameters) will be calculated and used in any derivation of summary
  statistics.
- Only planned assessment timepoints (according to Appendix 2: Schedule of Activities) will be included in data displays summarizing measurements by visit.
- Assessments not chosen for use in summary statistics will still appear in the associated listings.
- All applicable valid assessments, irrespective of proximity to the target study day, will be used when
  categorizing values across visits, such as 'maximum grade during the intervention phase' or 'at any time
  post-baseline', and for any algorithm that has specific rules for which observation to use (e.g. LOCF).

## **Change from Baseline**

- Post-Dose Visit Value Baseline
- Unless otherwise specified, the baseline definitions specified in Section 6.2 will be used for derivations for endpoints / parameters.

#### Study Day

- The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE) will be derived as the number of days between the date of the event and the Intervention Phase treatment start date as follows:
  - o If date of event ≥ start date of study treatment, then
    - Study Day = Date of Event Intervention Phase Treatment Start Date +1
  - If date of event < start date of study treatment, then</li>
    - Study Day = Date of Event Intervention Phase Treatment Start Date
  - Note that the start date of each phase is on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### Phase Day

 Calculated as the number of days from First Dose Date of CAB + RPV for the respective phase (based on study period classifications in <u>Table 3</u>):

#### OLI phase:

- If Assessment Date < First Dose Date of Oral CAB + RPV then
  - Phase Day = Assessment Date First Dose Date of Oral CAB + RPV
- If Assessment Date ≥ First Dose Date of Oral CAB + RPV then
  - Phase Day = Assessment Date First Dose Date of Oral CAB + RPV +1

#### Injection phase:

- If Assessment Date < Dose Date of Injection CAB + RPV then</li>
  - Phase Day = Assessment Date Dose Date of Injection CAB + RPV
- If Assessment Date ≥ Dose Date of Injection CAB +RPV then
  - Phase Day = Assessment Date Dose Date of Injection CAB + RPV +1

#### Follow-up phase:

- If Assessment Date < Follow-up Week 4 Visit Date then</li>
  - Phase Day = Assessment Date Follow-up Week 4 Visit Date
- If Assessment Date ≥ Follow-up Week 4 Visit Date then
  - Phase Day = Assessment Date Follow-up Week 4 Visit Date +1

## 11.5.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing day and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied. Consequently, the age
  of the subject will not be calculated and will remain missing.

#### **Body Mass Index (BMI)**

• Calculated in the CRF as Weight (kg) / [Height (m)<sup>2</sup>]

## 11.5.3. Safety

#### **Exposure**

#### Compliance

Compliance for the OLI Phase will be calculated as follows:

OLI Compliance 
$$\% = \frac{\# days \ subject \ took \ the \ study \ drug}{Minimum \ (\# \ of \ days \ subject \ was \ enrolled \ in \ the \ OLI \ period,28)}$$

#### **Extent of Exposure**

• Exposure to CAB+RPV Oral Lead-in = IP (oral lead-in) stop date - IP (oral lead-in) start date +1

#### **Duration (Days)**

• AE Resolution Date - AE Start Date + 1

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value. If a character value starting with "<=x", then the numeric value will be x.
  - Example 1: 2 Significant Digits = '< x 'becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' or '>=x' becomes x + 0.1

Example 3: 0 Significant Digits = '< x' becomes x – 1

#### 12-Lead Electrocardiograms

#### QTcB Interval

When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

If RR interval (in msec) is provided, then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{QT}{\sqrt{RR/1000}} \qquad QTcF = \frac{QT}{\sqrt[3]{RR/1000}}$$

where uncorrected QT interval is also measured in msec.

If RR interval is not provided directly and one of QTcB or QTcF has been entered, then RR interval can be obtained from the above formulas and used to calculate the other correction method value; i.e.,

$$QTcB = \sqrt{\frac{QTcF^{3}}{QT}}$$

$$QTcF = \sqrt[3]{QT \cdot QTcB^{2}}$$
#### 11.5.4. Pharmacokinetic

#### **Pharmacokinetic Parameter Statistics**

- For the purposes of calculating summary statistics and for statistical analysis, all PK parameters with the exception of t<sub>max</sub> will be log<sub>e</sub> transformed.
- Geometric coefficient of variation:
  - Untransformed Data: 100 \* (SD/Mean).
  - Transformed Data: 100 \* (sqrt(exp(SD<sub>log</sub><sup>2</sup>)-1)) where SD<sub>log</sub> indicates the standard deviation of logtransformed data

### 11.5.5. Health Outcomes





## 11.6. Appendix 6: Reporting Standards for Missing Data

## 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Withdrawn participants may be replaced in the study. All subjects who withdraw prematurely from the study/study drug will be documented and the reason for their withdrawal recorded in the final Clinical Pharmacology Study Report (CPSR).</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> <li>Withdrawal visits will be slotted according to Appendix 2: Assessment Windows</li> </ul> |

## 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| 0 " | . , |
| Outliers | <ul> <li>Any participants excluded from the summaries and/or statistical analyses will be<br/>documented along with the reason for exclusion in the clinical study report.</li> </ul> |
| CCI | Subjects who were injected that have missing ccl data may have it imputed with their last observation carried forward (LOCF) |

## 11.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in participant listing displays.</li> <li>Where necessary, partial dates may be imputed for specific analysis purposes as outlined below.</li> <li>Imputed partial dates will not be used to derive study day, time to onset or duration (e.g., time to onset or duration of AEs), or elapsed time variables (e.g., time since diagnosis).</li> </ul> |
| Adverse<br>Events | <ul> <li>Imputations in the AEs dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.</li> <li>Partial dates for AE recorded in the eCRF will be imputed using the following conventions:</li> </ul> |
| | <ul> <li>Missing start day</li> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> </ul> </li> </ul> |

| Element | Reporting Detail | |
|---|---|---|
| | | <ul> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing stop day | Last day of the month will be used. |
| | Missing stop day and month | No Imputation |
| | Completely missing start/end date | No imputation |
| Concomitant<br>Medications | | ng start or end dates will remain missing, with no imputation applied. any concomitant medications recorded in the eCRF will be imputed acconvention: |
| | doing are renewii | g contention. |
| | Missing start day | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year) |
| | Missing end day and month | A '31' will be used for the day and 'Dec' will be used for the month. |
| | Completely missing start/end date | No imputation |
| | The recorded part | tial date will be displayed in listings. |

## 11.7. Appendix 7: Values of Potential Clinical Importance

#### 11.7.1. Laboratory Values

Laboratory values will be graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1, March 2017, as specified in the protocol Appendix 11.7, and shown below:





### 11.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|----------|------------------------|-------|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | <320 | >450 |
| Absolute PR Interval | msec | <120 | >220 |
| Absolute QRS Interval | msec | <70 | >120 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

# 11.8. Appendix 8: Abbreviations & Trademarks

## 11.8.1. Abbreviations

| ADaM | Analysis data model |
|---|---|
| AE | Adverse event |
| ALT | alanine aminotransferase (SGPT) |
| AST | Aspartate aminotransferase (SGOT) |
| ATC | Anatomical Therapeutic Chemical Classification level |
| AUC <sub>0-t</sub> | Area under the concentration time curve from time zero to |
| 110 00-1 | last quantifiable time point |
| AUC <sub>0-τ</sub> | Area under the concentration-time curve over one dosing |
| 110 00 1 | interval |
| $AUC_{0-\infty}$ | Area under the concentration time curve from time zero to |
| | infinity |
| AUC <sub>0-24</sub> | Area under the concentration-time curve over 24 hours |
| BMI | Body mass index |
| BQL | Below the quantification limit |
| CAB | Cabotegravir |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence interval |
| C <sub>max</sub> | Maximum observed concentration |
| CPK | Creatine phosphokinase |
| CPMS | Clinical Pharmacokinetic Modelling Simulation |
| C24 | Concentration at 24-hour timepoint |
| Ст | Last observed quantifiable concentration |
| CV | Coefficient of variance |
| $CV_b$ | Geometric Coefficient of variation |
| ECG | Electrocardiogram |
| GSK | GlaxoSmithKline |
| HIV | Human immunodeficiency virus |
| НО | Health Outcomes |
| IDSL | Integrated Data Standards Library |
| IM | Intramuscular |
| IP | Investigational product |
| ISR | Injection site reaction |
| K <sub>A</sub> LA | Absorption rate constant, Long-acting |
| $\lambda_{\rm z}$ | Terminal phase rate constant |
| LA | Long-acting |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Mg | Milligrams |
| mL | Milliliter |
| NNRTI | Non-nucleoside reverse transcriptase inhibitor |
| NQ | Non-quantifiable |
| CCI | |

| OLI | Oral Lead In |
|---|---|
| PK | Pharmacokinetic(s) |
| CCI | |
| QTcB | QT duration corrected for heart rate by Bazett's formula |
| QTcF | QT duration corrected for heart rate by Fridericia's formula |
| RAP | Reporting and Analysis Plan |
| RPV | Rilpivirine |
| SAE | Serious adverse event(s) |
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| SoA | Schedule of Activities |
| SOP | Standard operating procedure |
| t <sub>1/2</sub> | Apparent terminal phase half-life |
| τ | Dosing interval |
| t <sub>max</sub> | Time of occurrence of Cmax |
| ULN | Upper limit of normal |

## 11.8.2. Trademarks

| Trademarks of ViiV Healthcare |
|-------------------------------|
| NONE |

| Trademarks not owned by ViiV<br>Healthcare |
|--------------------------------------------|
| MedDRA |
| SAS |
| Winnonlin |

## 11.9. Appendix 9: List of Data Displays

All data displays will use the term "subject" rather than "participant" in accordance with CDSIC and GSK Statistical Display Standards.

The list of data displays included in this critical component RAP is tentative, to be confirmed and modified as appropriate during the development of the full RAP.

### 11.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.10 | N/A |
| Safety | 3.1 to 3.37 | 3.38 |
| Pharmacokinetic | 4.1 to 4.4 | 4.5 to 4.10 |
| Health Outcomes | 6.1 to 6.7 | N/A |
| Section Listings | | ings |
| ICH Listings | 1 to 24 | |
| Other Listings | 25 to 38 | |

#### 11.9.2. Deliverables

| Delivery | Description |
|----------|-------------------------------------------------------------------|
| Interim | Informal Interim PK Analyses at Week 4 and Week 12 post injection |
| SAC | Final Statistical Analysis Complete |

# 11.9.3. Study Population Tables

| Study | Population Tab | les | | | 1 |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | Safety | DISP_T1 | Summary of Subject Disposition at Each Study Phase | ICH E3 | SAC |
| 1.3. | Safety | DISP_T2 | Summary of Reasons for Withdrawal at Each Study Phase | | SAC |
| 1.4. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| Protoc | ol Deviation | | | | |
| 1.5. | Safety | DV1 | Summary of Important Protocol Deviations by Study Phase and Overall | ICH E3 | SAC |
| Popula | tion Analysed | | | | |
| 1.6. | Enrolled | SP1 | Summary of Study Populations by Study Phase and Overall | GSK Statistical Display Standard Note: Show n's at each study phase. | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.7. | Safety | DM1 | Summary of Demographics and Baseline Characteristics | ICH E3, FDAAA, EudraCT<br>Note: To include Age Ranges | SAC |
| 1.8. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 1.9. | Safety | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC |
| 1.10. | Safety | CM1 | Summary of Concomitant Medications by Study Phase and Overall | ICH E3 | SAC |

# 11.9.4. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | ire and Treatmo | ent Compliance | | | |
| 3.1. | Safety | 207966/primary_15/<br>T3.1 | Summary of Exposure to Study Treatment | ICH E3 Display treatment in columns. Include the following parameters: "Exposure (Days-oral lead-in)" "Exposure (Weeks-oral lead-in)" "Oral Lead-in Compliance %" from 11.5.3 "No. of Subjects Receiving Injections" "Number of Injections" | SAC |
| Advers | e Events (AEs) | | | | |
| 3.2. | Safety | AE13 | Adverse Event Overview by Study Phase and Overall | High level summary to include counts of overall AEs, Treatment emergent AEs, Serious AEs, AEs leading to withdrawal, related AEs, serious related AEs, AEs related to Covid-19, AEs related to Covid-19 leading to withdrawal, fatal AEs Repeat for each study phase and overall | SAC |
| 3.3. | Safety | AE1xo | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.4. | Safety | AE5B | Summary of All Adverse Events by System Organ Class, Preferred Term, and Maximum Grade | ICH E3 Repeat for each study phase and overall | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.5. | Safety | AE15 | Summary of Common (>=10%) Adverse Events by Overall Frequency (Number of Subjects and Occurrences) | ICH E3 Note: "Common" AEs will be based on the Total column. Repeat for each study phase and overall | SAC |
| 3.6. | Safety | AE5B | Summary of Common (>=10%) Adverse Events by System Organ Class, Preferred Term, and Maximum Grade | ICH E3 Note: "Common" AEs will be based on the Total column. Repeat for each study phase and overall | SAC |
| 3.7. | Safety | AE5B | Summary of Drug-Related Adverse Events by System Organ Class, Preferred Term, and Maximum Grade | ICH E3 Repeat for each study phase and overall | SAC |
| 3.8. | Safety | AE15 | Summary of Common (>=10%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT Note: "Common" AEs will be based on the Total column. Repeat for each study phase and overall | SAC |
| Serious | and Other Sig | nificant Adverse Ev | ents | | |
| 3.9. | Safety | AE5B | Summary of Serious Adverse Events by System Organ Class, Preferred Term, and Maximum Grade | ICH E3 Repeat for each study phase and overall | SAC |
| 3.10. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT<br>Repeat for each study phase and<br>overall | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.11. | Safety | AE5B | Summary of Serious, Drug-Related Adverse Events by System Organ Class, Preferred Term, and Maximum Grade | Repeat for each study phase and overall | SAC |
| 3.12. | Safety | AE5B | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class, Preferred Term, and Maximum Grade | GSK Statistical Display Standard<br>Repeat for each study phase and<br>overall | SAC |
| 3.13. | Safety | AE5B | Summary of All Drug-Related Adverse Events Excluding Injection Site Reactions by System Organ Class, Preferred Term, and Maximum Grade | Repeat for each study phase and overall | SAC |
| 3.14. | Safety | PAN1A | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events | Note: To also include results of Covid-<br>19 tests performed | SAC |
| 3.15. | Safety | AE5B | Summary of Covid-19 Adverse Events by System Organ Class, Preferred Term, and Maximum Grade | Repeat for each study phase and overall | SAC |
| 3.16. | Safety | AE1xo | Summary of Covid-19 Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | Repeat for each study phase and overall | SAC |
| 3.17. | Safety | AE15 | Summary of Serious Covid-19 Adverse Events by System Organ Class, and Preferred Term (Number of Subjects and Occurrences) | Repeat for each study phase and overall | SAC |
| 3.18. | Safety | PAN3A | Summary of Covid-19 Symptoms for Subjects with COVID-19 Adverse Events | Note: data collected from AE_covid-19 eCRF | SAC |
| 3.19. | Safety | PAN10A | Incidence of Covid-19 Adverse Events by Gender and Pandemic Course | Pandemic course = During and Post pandemic Post pandemic date to be provided upon availability. | SAC |

| Injectio | n Site Reaction | n Adverse Events | | | |
|---|---|---|---|---|---|
| 3.20. | Safety | 201584/primary_7/T<br>3.43 | Summary of Subject-Level Characteristics of Injection Site Reaction Adverse Events by Treatment and Overall | Treatment to be listed in the columns | SAC |
| 3.21. | Safety | 201584/primary_7/T<br>3.40 | Summary of Injection Site Reaction Adverse Events (Event-<br>Level Summary) by Treatment and Overall | Treatment to be listed in the columns | SAC |
| 3.22. | Safety | 201584/primary_7/T<br>3.46 | Summary of Subject-Level Characteristics of Injection Site Reaction Adverse Events by Maximum Grade, Treatment, and Overall | Treatment to be listed in the columns | SAC |
| Advers | e Events of Sp | ecial Interest | | | |
| 3.23. | Safety | 201584/primary_07/<br>T3.134 | Summary of Seizure Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 3.24. | Safety | 201584/primary_07/<br>T3.137 | Summary of Hepatic Safety Profile: Assessment of Risk of Hepatotoxicity Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| Laborat | tory: Chemistr | y | | | |
| 3.25. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Study Phase and Visit | ICH E3 | SAC |
| 3.26. | Safety | LB1 | Summary of Chemistry Values by Study Phase and Visit | ICH E3 | SAC |
| 3.27. | Safety | LB16 | Summary of Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 Repeat for each study phase | SAC |
| Laborat | tory: Hematolo | gy | | | |
| 3.28. | Safety | LB1 | Summary of Hematology Changes from Baseline by Study Phase and Visit | ICH E3 | SAC |
| 3.29. | Safety | LB1 | Summary of Hematology Values by Study Phase and Visit | ICH E3 | SAC |
| 3.30. | Safety | LB16 | Summary of Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 Repeat for each study phase | SAC |

| Laborat | tory: Urinalysis | 3 | | | |
|---|---|---|---|---|---|
| 3.31. | Safety | UR1 | Summary of Worst-Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline by Study Phase | ICH E3 Note: Define change categories according to actual values expected from lab dataset Repeat for each study phase and overall | SAC |
| Laborat | tory: Hepatobil | iary (Liver) | | | |
| 3.32. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting by Study Phase and Overall | GSK Statistical Display Standard Note: See Appendix 11.4.4 for Criteria | SAC |
| 3.33. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities by Study Phase and Overall | GSK Statistical Display Standard Note: See Appendix 11.4.4 for Criteria | SAC |
| ECG | | | | | |
| 3.34. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Study Phase and Visit | GSK Statistical Display Standard | SAC |
| 3.35. | Safety | EG2 | Summary of ECG Values by Study Phase and Visit | GSK Statistical Display Standard | SAC |
| 3.36. | Safety | EG1 | Summary of ECG Findings by Study Phase and Visit | GSK Statistical Display Standard | SAC |
| Vital Sig | /ital Signs | | | | |
| 3.37. | Safety | VS1 | Summary of Change from Baseline in Vital Signs by Study Phase and Visit | ICH E3 | SAC |

# 11.9.5. Safety Figures

| Safety | Safety Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 3.38. | Safety | AE10 | Plot of Common (>=10%) Adverse Events by Relative Risk, Study Phase, and Overall | Note: Display a different plot for each phase and overall | SAC |

## 11.9.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic Parar | neters | | | |
| 4.1. | PK<br>Parameter | PK_01 | Summary of Derived Plasma Cabotegravir PK Parameters by Study Phase | | Interim, SAC |
| 4.2. | PK<br>Parameter | PK_01 | Summary of Derived Plasma Rilpivirine PK Parameters by Study Phase | | Interim, SAC |
| Pharma | acokinetic Conc | entration | | | |
| 4.3. | PK<br>Concentration | PK01 | Summary of Plasma Cabotegravir PK Concentration (ug/mL)-<br>Time Data by Study Phase and Nominal Timepoint | | SAC |
| 4.4. | PK<br>Concentration | PK01 | Summary of Plasma Rilpivirine PK Concentration (ng/mL)-Time Data by Study Phase and Nominal Timepoint | | SAC |

# 11.9.7. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic Mea | n/Median Plots | | | |
| 4.5. | PK<br>Parameter | PK17 | Mean (SD) Plasma Cabotegravir Concentration-Time Plots (Linear and Semi-Log) by Study Phase | Display oral and LA phases on separate pages | SAC |
| 4.6. | PK<br>Parameter | PK17 | Mean (SD) Plasma Rilpivirine Concentration-Time Plots (Linear and Semi-Log) by Study Phase | Display oral and LA phases on separate pages | SAC |
| 4.7. | PK<br>Parameter | PK20 | Median (5 <sup>th</sup> and 95 <sup>th</sup> Percentile) Plasma Cabotegravir<br>Concentration-Time Plots (Linear and Semi-Log) by Study<br>Phase | Display oral and LA phases on separate pages | SAC |
| 4.8. | PK<br>Parameter | PK20 | Median (5 <sup>th</sup> and 95 <sup>th</sup> Percentile) Plasma Rilpivirine<br>Concentration-Time Plots (Linear and Semi-Log) by Study<br>Phase | Display oral and LA phases on separate pages | SAC |
| Pharma | acokinetic Indi | vidual Subject Plo | ots | | |
| 4.9. | PK<br>Parameter | PK16a | Individual Plasma Cabotegravir Concentration-Time Plots (Linear and Semi-Log) by Study Phase | Display oral and LA phases on separate pages | SAC |
| 4.10. | PK<br>Parameter | PK16a | Individual Plasma Rilpivirine Concentration-Time Plots (Linear and Semi-Log) by Study Phase | Display oral and LA phases on separate pages | SAC |

### 11.9.8. Health Outcomes Tables

| Health | lealth Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Quest | tionnaire Outc | omes | | | |
| 6.1. | Safety | 201584/primary_07/T6.2 | CCI | | SAC |
| 6.2. | Safety | 201584/primary_07/T6.1 | | | SAC |
| 6.3. | Safety | 201584/primary_07/T6.35 | | | SAC |
| 6.4. | Safety | 201584/primary_07/T6.36 | | | SAC |
| 6.5. | Safety | 201584/primary_07/T6.37 | | | SAC |
| 6.6. | Safety | 201584/primary_07/T6.38 | | | SAC |
| 6.7. | Safety | 201584/primary_07/T6.39 | | | SAC |

# 11.9.9. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 2. | Screened | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| Protoc | ol Deviations | | | | |
| 3. | Screened | DV2 | Listing of Protocol Deviations | ICH E3 Note: Include flag for important deviations (Y/N) and Covid-19 relatedness (Y/N) | SAC |
| 4. | Screened | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 5. | Screened | SP3 | Listing of Subjects Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 6. | Screened | DM2 | Listing of Demographic Characteristics | ICH E3 Include column indicating inclusion in the enrolled (Y/N) and safety populations (Y/N) | SAC |
| 7. | Screened | DM9 | Listing of Race | ICH E3 Include column indicating inclusion in the enrolled (Y/N) and safety populations (Y/N) | SAC |
| Exposi | ure and Treatm | ent Compliance | | | |
| 8. | Screened | EX3 | Listing of Exposure Data | ICH E3 | SAC |

| Advers | se Events | | | | |
|---|---|---|---|---|---|
| 9. | Screened | AECP | Listing of All Adverse Events | ICH E3 Include column indicating Phase | SAC |
| 10. | Screened | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 Replace the column for treatment with Phase | SAC |
| 11. | Screened | AECP | Listing of Serious Adverse Events | ICH E3 Include column indicating Phase Note: Include Fatal vs Non-Fatal Designation | SAC |
| 12. | Screened | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 13. | Screened | AECP | Listing of Adverse Events Leading to Withdrawal from Study or<br>Permanent Discontinuation of Study Treatment | ICH E3 Include column indicating Phase | SAC |
| 14. | Screened | AECP | Listing of Covid-19 Adverse Events | ICH E3 Include column indicating Phase Note: Display Covid-19 Adverse events and descriptive details | SAC |
| 15. | Screened | PAN12 | Listing of COVID-19 Assessments and Symptom Assessments | | SAC |
| 16. | Screened | PAN5 | Listing of Dates of COVID-19 Pandemic Measures | Include Pandemic End date if available | SAC |
| All Lab | oratory | | | | |
| 17. | Screened | LB5 | Listing of Continuous Laboratory Data by Lab Category, Study Phase, and Visit | ICH E3 Note: Include Chemistry and Hematology results | SAC |
| 18. | Screened | LB14 | Listing of Categorical Laboratory Data by Lab Category, Study Phase, and Visit | ICH E3 Note: Include Urinalysis, Coagulation, Drugs, and Infectious Disease results | SAC |
| 19. | Screened | EG3 | Listing of ECG Values by Study Phase and Visit | Sort by Phase and Visit | SAC |
| 20. | Screened | EG5 | Listing of ECG Findings by Study Phase and Visit | Sort by Phase and Visit | SAC |
| 21. | Screened | VS4 | Listing of Vital Signs by Study Phase and Visit | Sort by Phase and Visit | SAC |

| 22. | Screened | PREG1 | Listing of Subjects Who Became Pregnant During the Study | SAC |
|---|---|---|---|---|
| PK | | | | |
| 23. | Screened | PK07 | Listing of Plasma Cabotegravir PK Concentration-Time Data by study phase | SAC |
| 24. | Screened | PK07 | Listing of Plasma Rilpivirine PK Concentration-Time Data by study phase | SAC |

# 11.9.10. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display<br>Standard / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 25. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 26. | Screened | SD2 | Listing of End of Study Record for Subjects Affected by Covid-19 | Covid-19 relatedness as determined by Covid related AEs, PDs, missed visits, & Disposition | SAC |
| Prior an | d Concomitan | nt Medications | | | |
| 27. | Screened | MH2 | Listing of Medical History for All Subjects | | SAC |
| 28. | Screened | CM3 | Listing of Prior Medications | GSK Statistical Display Standard | SAC |
| 29. | Screened | CM3 | Listing of Concomitant Medications by Study Phase | GSK Statistical Display Standard | SAC |
| Adverse | e Events | | | | |
| 30. | Screened | AE8 | Listing of Injection Site Reaction Adverse Events | | SAC |
| 31. | Screened | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | GSK Statistical Display Standard | SAC |
| Laborat | Laboratory Results | | | | |
| 32. | Screened | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | Note: See Appendix 11.4.4 for Criteria | SAC |
| 33. | Screened | LIVER13 | Listing Subjects Meeting Hepatobiliary Lab Abnormality Criteria | Note: See Appendix 11.4.4 for Criteria | SAC |

| PK | | | | |
|---|---|---|---|---|
| 34. | Screened | PK13 | Listing of Derived Plasma Cabotegravir PK Parameters by study phase | SAC |
| 35. | Screened | PK13 | Listing of Derived Plasma Rilpivirine PK Parameters by study phase | |
| Health ( | Outcome | | | |
| 36. | Screened | HO_01 | Listing of CCI Scores | SAC |
| 37. | Screened | HO_02 | Listing of CCI Questionnaire Results at Day 8 | SAC |
| 38. | Screened | HO_03 | Listing of CCI from Daily Diary Cards | SAC |

## 11.9.11. Mock Displays

Protocol: 208832 

Population: Safety

Table DISP\_T1
Summary of Subject Disposition at Each Study Phase

| Study Phase | | Total (N=200) |
|--------------------|---------------------|---------------|
| | | 4 01 |
| Oral Lead-in Phase | ENTERED | xx (xx.x%) |
| | COMPLETED | xx (xx.x%) |
| | WITHDRAWN | xx (xx.x%) |
| | COVID-19 RELATED[1] | xx (xx.x%) |
| Injection Phase | ENTERED | xx (xx.x%) |
| | COMPLETED | xx (xx.x%) |
| | WITHDRAWN | xx (xx.x%) |
| | COVID-19 RELATED[1] | xx (xx.x%) |
| Follow-up Phase | ENTERED | xx (xx.x%) |
| | COMPLETED | xx (xx.x%) |
| | WITHDRAWN | xx (xx.x%) |
| | COVID-19 RELATED[1] | xx (xx.x%) |

<sup>[1]</sup> Covid-19 Related Disposition as collected from the Study Impact record

208832

Protocol: 208832 

[1]

Population: Safety

Table DISP\_T2 Summary of Reasons for Withdrawal at Each Study Phase

| Primary Reason | Oral CAB 30mg<br>+ Oral RPV<br>25mg (N=100) | IM CAB 600mg<br>+ IM RPV<br>900mg -<br>Injection<br>Phase<br>(N=100) | IM CAB 600mg + IM RPV 900mg - Follow-up Phase (N=100) | Overall<br>(N=100) |
|---|---|---|---|---|
| ADVERSE EVENT | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 RELATED[1] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x = (xx.x%) |
| PROTOCOL DEVIATION | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 RELATED[1] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x = (xx.x%) |
| SUBJECT REACHED PROTOCOL-DEFINED STOPPING | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| CRITERIA | | | | |
| STUDY TERMINATED BY SPONSOR | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| LOST TO FOLLOW-UP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| INVESTIGATOR SITE CLOSED | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PHYSICIAN DECISION | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| WITHDRAWAL BY SUBJECT | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| COVID-19 RELATED[1] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

Covid-19 Related Disposition as collected from the Study Impact record

Protocol: 208832 Page 1 of x

Population: Pharmacokinetic Parameter

 $$\rm PK\_01$$  Summary of Derived Cabotegravir Pharmacokinetic Parameters by Phase

| Parameter | Summary Statistics | Oral CAB 30mg<br>(N=xx) | IM CAB 600 mg (N=xx) |
|---|---|---|---|
| AUC <sub>0-t</sub> (h*μg/mL) | n | xx | xx |
| | Mean (SD) | Xxx.x (xx.xx) | Xxx.x (xx.xx) |
| | 95% CI | (xxx.xx,xxx) | (xxx.xx,xxx.xx) |
| | %CV | XX.X | XX.X |
| | Median | | |
| | | xxx.xx | xxx.xx |
| | Min, Max | XXX.X, XXX.X | XXX.X, XXX.X |
| | Geometric mean | xxx.xx | xxx.xx |
| | 95% CI | (xxx.xxx,xxx.xxx) | (xxx.xxx,xxx.xxx) |
| | SD (log) | xxx.xxx | xxx.xxx |
| | Geometric %CV | xxx.x | xxx.x |
| AUC <sub>0-∞</sub> (h*μg/mL) | n | xx | xx |
| | Mean (SD) | Xxx.x (xx.xx) | Xxx.x (xx.xx) |
| | 95% CI | (xxx.xx,xxx.xx) | (xxx.xx,xxx.xx) |
| | %CV | xx.x | xx.x |
| | Median | xxx.xx | xxx.xx |
| | Min, Max | xxx.x, xxx.x | xxx.x, xxx.x |
| | Geometric mean | xxx.xx | xxx.xx |
| | 95% CI | (xxx.xxx,xxx.xxx) | (xxx.xxx,xxx.xxx) |
| | SD (log) | xxx.xxx | xxx.xxx |

208832

XXX.X

xxx.x

/Directory/program.sas 01JAN2002 12:01

Geometric %CV

### Programming notes:

- 1) Repeat table for RPV (Oral RPV 25mg, IM RPV 900mg; ng/mL, ng\*h/mL)
- 2) Repeat for all of the following PK parameters as available: C<sub>max</sub>, t<sub>max</sub>, t<sub>1/2</sub>, K<sub>A</sub> LA, λz, C24, Cτ
- 3) For t<sub>max</sub>, only the n, median, minimum, and maximum should be provided.
- 4) Report the means & median +1 decimal past the maximum length of results within parameter. Report the SD and 95% CI values +2 decimals past the maximum length of results within parameter. %CV statistics should be reported to 1 decimal.

Protocol: 208832 

Population: Screened

| | Listing of CO | HO 01 | Score | es |
|---|---|---|---|---|
| Treatment | Site Id./<br>Unique Subject Id. | Treatment/<br>Injection Site<br>Side | Visit | Date CCI |
| Treatment A | PPD | CAB/Left | Day 1 | YYYY-MM-DDTHH:MM |
| | | | Day 2 | YYYY-MM-DDTHH:MM |
| | | | Day 4 | YYYY-MM-DDTHH:MM |
| | | | Day 5 | YYYY-MM-DDTHH:MM |
| | | | Day 8 | YYYY-MM-DDTHH:MM |
| | | RPV/Right | Day 1 | YYYY-MM-DDTHH:MM |

USER ID:/PROGRAM PATH/PROGRAM DATE TIME

208832

Protocol: 208832 
Population: Screened

HO 02
Listing of Results at Day 8

Treatment: Treatment A



. . .

YYYY-MM-DD/ RPV/Right HH:MM

CC

CC

USER ID:/PROGRAM PATH/PROGRAM DATE TIME

Protocol: 208832 

Population: Screened

HO\_03
Listing of Injection Area Symptoms from Daily Diary Cards

| Treatment | Site Id./<br>Unique Subject Id. | _ | Assessment/ | Symptoms? (Y/N) | Pain<br>(0-3) | Itching (0-3) | | Home<br>Treatment [2] |
|---|---|---|---|---|---|---|---|---|
| Treatment A | PPD | CAB/<br>Left | YYYY-MM-DD/ | Y | 2 | 1 | BU, SF | AP, Top |
| | | | YYYY-MM-DD/<br>2 | Y | 0 | 1 | | Тор |
| | | RPV/<br>Right | YYYY-MM-DD/<br>1 | N | | | | |

USER ID:/PROGRAM PATH/PROGRAM DATE TIME

<sup>[1]</sup> NO=None, BR=Bruising, BU=Bump, D=Discoloration, R=Redness, SF=Skin firmness, SW=Swelling, W=Warm to touch. [2] NO=None, AP=Acetaminophen/paracetamol (Tylenol), D=Diphenhydramine (Benadryl), Top=Topical anti-itch cream or ointment such as hydrocortisone/diphenhydramine, etc., W=Warm compress (heating pad), C=Cold compress (cold pack or ice pack).

# 11.10. Appendix 10: AESI Identification

SMQ and PT codes based on MedDRA dictionary version 23.0.

## 11.10.1. Hepatotoxicity

| SMQ: Hepatic failure, fibrosis and cirrhosis and other liver damage-<br>related conditions<br>SMQ Code: 20000013<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cardiohepatic syndrome | 10082480 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10072268 |
| Duodenal varices | 10051010 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |

| Gastric varices haemorrhage | 10057572 |
|----------------------------------------------------|----------|
| Gastrooesophageal variceal haemorrhage prophylaxis | 10066597 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |
| Immune-mediated cholangitis | 10083406 |
| Immune-mediated hepatic disorder | 10083521 |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Liver dialysis | 10076640 |

| Liver disorder | 10024670 |
|---------------------------------------|----------|
| Liver injury | 10067125 |
| | 10067123 |
| Liver operation | |
| Liver transplant | 10024714 |
| Lupoid hepatic cirrhosis | 10025129 |
| Minimal hepatic encephalopathy | 10076204 |
| Mixed liver injury | 10066758 |
| Nodular regenerative hyperplasia | 10051081 |
| Nonalcoholic fatty liver disease | 10082249 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices | 10073215 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |

| | 1000000 |
|---|---|
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Sugiura procedure | 10083010 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |
| SMQ: Hepatitis, non-infectious<br>SMQ Code: 20000010<br>Category: A<br>Scope: Narrow | |
| Preferred Term | PT Code |
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |
| Non-alcoholic steatohepatitis | 10053219 |
| | · |

| Radiation hepatitis | 10051015 |
|---------------------|----------|
| Steatohepatitis | 10076331 |

# 11.10.2. Seizures

| SMQ: 'Convulsions'<br>SMQ Code: 20000079<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| 1p36 deletion syndrome | 10082398 |
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Alpers disease | 10083857 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| CEC syndrome | 10083749 |
| CDKL5 deficiency disorder | 10083005 |
| Change in seizure presentation | 10075606 |
| Clonic convulsion | 10053398 |
| Congenital bilateral perisylvian syndrome | 10082716 |

| Convulsive threshold lowered CSWS syndrome 10078827 Deja vu 10012177 Double cortex syndrome 10073490 Dreamy state 10013634 Drug withdrawal convulsions 10013752 Early infantile epileptic encephalopathy with burst-suppression 10071545 Eclampsia 10014129 Epilepsy 10015037 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079424 Frontal lobe epilepsy Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10078727 GM2 gangliosidosis Grey matter heterotopia Hemimegalencephaly Hyperglycaemic seizure 10071394 | Convulsion in childhood | 10052391 |
|---|---|---|
| CSWS syndrome 10078827 Deja vu 10012177 Double cortex syndrome 10073490 Dreamy state 10013634 Drug withdrawal convulsions 10013752 Early infantile epileptic encephalopathy with burst-suppression 10071545 Eclampsia 10014129 Epilepsy 10015037 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onic-clonic seizure 10083376 Generalised tonic-clonic seizure 10078100 Glucose transporter type 1 deficiency syndrome 10078100 Grey matter heterotopia 10082084 Hemimegalencephaly 10071394 Hyperglycaemic seizure 10071394 | Convulsions local | 10010920 |
| Deja vu 10012177 Double cortex syndrome 10073490 Dreamy state 10013634 Drug withdrawal convulsions 10013752 Early infantile epileptic encephalopathy with burst-suppression 10071545 Eclampsia 10014129 Epilepsy 10015037 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10083376 Generalised tonic-clonic seizure 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Convulsive threshold lowered | 10010927 |
| Double cortex syndrome Dreamy state Dreamy state Dreamy state Drug withdrawal convulsions 10013752 Early infantile epileptic encephalopathy with burst-suppression Eclampsia 10014129 Epilepsy 10015037 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10082084 Hemimegalencephaly Hyperglycaemic seizure 10071394 | CSWS syndrome | 10078827 |
| Dreamy state 10013634 Drug withdrawal convulsions 10013752 Early infantile epileptic encephalopathy with burst-suppression 10071545 Eclampsia 10014129 Epilepsy 10015037 Epilepsy 10079824 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10082084 Hemimegalencephaly 10071394 | Deja vu | 10012177 |
| Drug withdrawal convulsions Early infantile epileptic encephalopathy with burst-suppression Eclampsia 10014129 Epilepsy 10015037 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis Grey matter heterotopia Hyperglycaemic seizure 10071394 | Double cortex syndrome | 10073490 |
| Early infantile epileptic encephalopathy with burst-suppression Eclampsia 10014129 Epilepsy 10015037 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis Grey matter heterotopia Hyperglycaemic seizure 10071394 | Dreamy state | 10013634 |
| Eclampsia 10014129 Epilepsy 10015037 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Drug withdrawal convulsions | 10013752 |
| Epilepsy Union 10015037 Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Early infantile epileptic encephalopathy with burst-suppression | 10071545 |
| Epilepsy surgery 10079824 Epilepsy with myoclonic-atonic seizures 10081179 Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Eclampsia | 10014129 |
| Epilepsy with myoclonic-atonic seizures Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10082084 Hemimegalencephaly Hyperglycaemic seizure 10071394 | Epilepsy | 10015037 |
| Epileptic aura 10015049 Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Epilepsy surgery | 10079824 |
| Epileptic psychosis 10059232 Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10082084 Hemimegalencephaly 10078100 Hyperglycaemic seizure 10071394 | Epilepsy with myoclonic-atonic seizures | 10081179 |
| Febrile convulsion 10016284 Febrile infection-related epilepsy syndrome 10079438 Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Epileptic aura | 10015049 |
| Febrile infection-related epilepsy syndrome Focal dyscognitive seizures Frontal lobe epilepsy Gelastic seizure 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Epileptic psychosis | 10059232 |
| Focal dyscognitive seizures 10079424 Frontal lobe epilepsy 10049424 Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Febrile convulsion | 10016284 |
| Frontal lobe epilepsy Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Febrile infection-related epilepsy syndrome | 10079438 |
| Gelastic seizure 10082918 Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10078100 Hyperglycaemic seizure 10071394 | Focal dyscognitive seizures | 10079424 |
| Generalised onset non-motor seizure 10083376 Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10082084 Hemimegalencephaly 10078100 Hyperglycaemic seizure 10071394 | Frontal lobe epilepsy | 10049424 |
| Generalised tonic-clonic seizure 10018100 Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10082084 Hemimegalencephaly 10078100 Hyperglycaemic seizure 10071394 | Gelastic seizure | 10082918 |
| Glucose transporter type 1 deficiency syndrome 10078727 GM2 gangliosidosis 10083933 Grey matter heterotopia 10082084 Hemimegalencephaly 10078100 Hyperglycaemic seizure | Generalised onset non-motor seizure | 10083376 |
| GM2 gangliosidosis 10083933 Grey matter heterotopia 10082084 Hemimegalencephaly 10078100 Hyperglycaemic seizure 10071394 | Generalised tonic-clonic seizure | 10018100 |
| Grey matter heterotopia 10082084 Hemimegalencephaly 10078100 Hyperglycaemic seizure 10071394 | Glucose transporter type 1 deficiency syndrome | 10078727 |
| Hemimegalencephaly 10078100 Hyperglycaemic seizure 10071394 | GM2 gangliosidosis | 10083933 |
| Hyperglycaemic seizure 10071394 | Grey matter heterotopia | 10082084 |
| | Hemimegalencephaly | 10078100 |
| Hypocalcaemic seizure 10072456 | Hyperglycaemic seizure | 10071394 |
| 71 | Hypocalcaemic seizure | 10072456 |

| Hyponatraemic seizure 10073183 Idiopathic generalised epilepsy 10071081 Infantile spasms 10021750 Juvenile myoclonic epilepsy 10071082 Lafora's myoclonic epilepsy 10054030 Lennox-Gastaut syndrome 10048816 Migraine-triggered seizure 10076676 Molybdenum cofactor deficiency 10069687 Multiple subpial transection 10079825 Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10082068 Neonatal epileptic seizure 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke esizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure anoxic 10039907 Seizure cluster 10031350 < | Hypoglycaemic seizure | 10048803 |
|---|---|---|
| Infantile spasms 10021750 Juvenile myoclonic epilepsy 10071082 Lafora's myoclonic epilepsy 10054030 Lennox-Gastaut syndrome 10048816 Migraine-triggered seizure 10076676 Molybdenum cofactor deficiency 10069687 Multiple subpial transection 10079825 Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Nconatal seizures 10082067 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076981 Post stroke seizure 10076981 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 | Hyponatraemic seizure | 10073183 |
| Juvenile myoclonic epilepsy 10071082 Lafora's myoclonic epilepsy 10054030 Lennox-Gastaut syndrome 10048816 Migraine-triggered seizure 10076676 Molybdenum cofactor deficiency 10069687 Multiple subpial transection 10079825 Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Nconatal scizures 10082067 Partial scizures 10061334 Partial scizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Idiopathic generalised epilepsy | 10071081 |
| Lafora's myoclonic epilepsy 10054030 Lennox-Gastaut syndrome 10048816 Migraine-triggered seizure 10076676 Molybdenum cofactor deficiency 10069687 Multiple subpial transection 10079825 Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Neonatal seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076981 Post stroke seizure 10076981 Postictal headache 10052470 Postictal pyschosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073990 Seizure 10039906 Seizure anoxic 10039907 | Infantile spasms | 10021750 |
| Lennox-Gastaut syndrome 10048816 Migraine-triggered seizure 10076676 Molybdenum cofactor deficiency 10069687 Multiple subpial transection 10079825 Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Neonatal seizures 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal state 10070669 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Juvenile myoclonic epilepsy | 10071082 |
| Migraine-triggered seizure 10076676 Molybdenum cofactor deficiency 10069687 Multiple subpial transection 10079825 Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Neonatal seizures 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal state 100748727 Postictal state 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Lafora's myoclonic epilepsy | 10054030 |
| Molybdenum cofactor deficiency 10069687 Multiple subpial transection 10079825 Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Neonatal seizure 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Lennox-Gastaut syndrome | 10048816 |
| Multiple subpial transection 10079825 Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Neonatal seizure 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Migraine-triggered seizure | 10076676 |
| Myoclonic epilepsy 10054859 Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Neonatal seizure 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Molybdenum cofactor deficiency | 10069687 |
| Myoclonic epilepsy and ragged-red fibres 10069825 Neonatal epileptic seizure 10082068 Neonatal seizures 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Multiple subpial transection | 10079825 |
| Neonatal epileptic seizure 10082068 Neonatal seizure 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Myoclonic epilepsy | 10054859 |
| Neonatal seizure 10082067 Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Myoclonic epilepsy and ragged-red fibres | 10069825 |
| Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10072469 Postictal psychosis 10070669 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Neonatal epileptic seizure | 10082068 |
| Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10039906 Seizure 10039907 | Neonatal seizure | 10082067 |
| Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10039906 Seizure 10039907 | Partial seizures | 10061334 |
| Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Partial seizures with secondary generalisation | 10056209 |
| Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Petit mal epilepsy | 10034759 |
| Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Polymicrogyria | 10073489 |
| Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Post stroke epilepsy | 10076982 |
| Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Post stroke seizure | 10076981 |
| Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Postictal headache | 10052470 |
| Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Postictal paralysis | 10052469 |
| Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Postictal psychosis | 10070669 |
| Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 | Postictal state | 10048727 |
| Seizure 10039906 Seizure anoxic 10039907 | Post-traumatic epilepsy | 10036312 |
| Seizure anoxic 10039907 | Schizencephaly | 10073487 |
| | Seizure | 10039906 |
| Seizure cluster 10071350 | Seizure anoxic | 10039907 |
| | Seizure cluster | 10071350 |

| Seizure like phenomena | 10071048 |
|---|---|
| Severe myoclonic epilepsy of infancy | 10073677 |
| Simple partial seizures | 10040703 |
| Status epilepticus | 10041962 |
| Sudden unexplained death in epilepsy | 10063894 |
| Temporal lobe epilepsy | 10043209 |
| Tonic clonic movements | 10051171 |
| Tonic convulsion | 10043994 |
| Tonic posturing | 10075125 |
| Topectomy | 10073488 |
| Transient epileptic amnesia | 10081728 |
| Tuberous sclerosis complex | 10080584 |
| Uncinate fits | 10045476 |
| Additional selected preferred terms from HLT "Disturbances in consciousness NEC" (Code: 10013509) under SOC "Nervous systems disorders" and HLT "Confusion and disorientation" (Code: 10010301) under SOC "Psychiatric disorders". | |
| Preferred Term | PT Code |
| Confusional state | 10010305 |
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10050093 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |

## 11.10.3. Torsade de pointes/QT prolongation

Notes: Medical concept of QT prolongation and complications. Only narrow terms from SMQ 'Torsade de pointes/QT prolongation' selected plus one additional PT under HLT 'ECG investigations'.

| SMQ: Torsade de pointes/QT prolongation<br>SMQ Code: 20000001<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Electrocardiogram QT interval abnormal | 10063748 |
| Electrocardiogram QT prolonged | 10014387 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Torsade de pointes | 10044066 |
| Ventricular tachycardia | 10047302 |
| Additional preferred terms selected from HLT ' ECG investigations' (Code: 10053104) under SOC 'Investigations'. | |
| Preferred Term | PT Code |
| Electrocardiogram repolarisation abnormality | 10052464 |

#### 11.10.4. COVID-19 Adverse Events

COVID-19 adverse events are identified based on MedDRA coded values and/or AE referenced in the COVID-19 Coronavirus Infection assessment. The Lowest Level Terms (LLTs) and codes, Preferred Terms (PTs), High Level Terms (HLTs), High Level Group Terms (HLGTs), and System Organ Classes (SOCs), below are from MedDRA 23.0. In case there is a change to the version of MedDRA at time of reporting, the coded values based on the MedDRA version at the time of reporting will be used. The additional events may also be added based on the blinded review of AE data collected on study prior to the database freeze.

SOC: Infections and infestations

| LLT code | LLT | PT | HLT | HLGT |
|---|---|---|---|---|
| | | Asymptomatic | Coronavirus | Viral infectious |
| 10084459 | Asymptomatic COVID-19 | COVID-19 | infections | disorders |

#### 

| LLT code | LLT | PT | HLT | HLGT |
|---|---|---|---|---|
| | Asymptomatic SARS- | Asymptomatic | Coronavirus | Viral infectious |
| 10084467 | CoV-2 infection | COVID-19 | infections | disorders |
| | | Coronavirus | Coronavirus | Viral infectious |
| 10053983 | Corona virus infection | infection | infections | disorders |
| | | Coronavirus | Coronavirus | Viral infectious |
| 10051905 | Coronavirus infection | infection | infections | disorders |
| | Coronavirus disease | | Coronavirus | Viral infectious |
| 10084382 | 2019 | COVID-19 | infections | disorders |
| | | | | Microbiology and |
| 10070255 | | Coronavirus | Virus identification | serology |
| | Coronavirus test positive | test positive | and serology | investigations |

#### 

| | | | | Thereneutie |
|---|---|---|---|---|
| | | | | Therapeutic |
| | | 00) (10, 40 | A (" C (' | procedures and |
| 10084460 | 00)//0 404 | COVID-19 | Antiinfective | supportive care |
| | COVID-19 treatment | treatment | therapies | NEC |
| 10084639 | | SARS-CoV-2 | Coronavirus | Viral infectious |
| | SARS-CoV-2 sepsis | sepsis | infections | disorders |
| | | | | Microbiology and |
| 10084271 | SARS-CoV-2 test | SARS-CoV-2 | Virus identification | serology |
| | positive | test positive | and serology | investigations |
| 10084640 | | SARS CoV-2 | Coronavirus | Viral infectious |
| | SARS CoV-2 viraemia | viraemia | infections | disorders |
| | | | Coronavirus | Viral infectious |
| 10084268 | COVID-19 | COVID-19 | infections | disorders |
| | COVID-19 respiratory | | Coronavirus | Viral infectious |
| 10084401 | infection | COVID-19 | infections | disorders |
| | SARS-CoV-2 acute | | Coronavirus | Viral infectious |
| 10084270 | respiratory disease | COVID-19 | infections | disorders |
| | | | Coronavirus | Viral infectious |
| 10084272 | SARS-CoV-2 infection | COVID-19 | infections | disorders |
| | | COVID-19 | Coronavirus | Viral infectious |
| 10084381 | Coronavirus pneumonia | pneumonia | infections | disorders |
| | · | COVID-19 | Coronavirus | Viral infectious |
| 10084380 | COVID-19 pneumonia | pneumonia | infections | disorders |
| | Novel COVID-19- | COVID-19 | Coronavirus | Viral infectious |
| 10084383 | infected pneumonia | pneumonia | infections | disorders |
| | 1 | Suspected | Coronavirus | Viral infectious |
| 10084451 | Suspected COVID-19 | COVID-19 | infections | disorders |
| | Suspected SARS-CoV-2 | Suspected | Coronavirus | Viral infectious |
| 10084452 | infection | COVID-19 | infections | disorders |
| | | SARS-CoV-2 | Infectious | Ancillary infectious |
| 10084461 | SARS-CoV-2 carrier | carrier | disorders carrier | topics |